# A Phase 3, Multicenter Study to Assess the Long Term Safety and Tolerability of ALKS 3831 in Subjects with Schizophrenia

**Unique Protocol ID:** ALK3831-A306

NCT Number: NCT02669758

**EudraCT Number:** 2015-003880-13

**Date of Protocol:** 25 April 2017



## CLINICAL STUDY PROTOCOL

#### ALK3831-A306

EudraCT Number: 2015-003880-13

Study title: A Phase 3, Multicenter Study to Assess the Long Term

Safety and Tolerability of ALKS 3831 in Subjects with

Schizophrenia

Document date: v 3.0 (incorporates Amendment 2.0): 25 Apr 2017

v 2.0 (incorporates Amendment 1.0): 28 Mar 2016

Original Protocol: 24 Sep 2015

Sponsor: Alkermes, Inc.

852 Winter Street Waltham, MA 02451

**USA** 

#### CONFIDENTIAL

Information and data in this protocol contain trade secrets and privileged or confidential information, which is the property of Alkermes, Inc. No person is authorized to make it public without the written permission of Alkermes, Inc. These restrictions or disclosures will apply equally to all future information supplied to you that is indicated as privileged or confidential.

# **CONTACT INFORMATION**

**Table 1:** Study Contact Information

| Role in Study | Name | Address and Telephone |
|---|---|---|
| Alkermes Medical Monitor | PPD | Alkermes Pharma Ireland, Ltd. |
| | | Connaught House |
| | | 1 Burlington Road |
| | | Dublin 4, Ireland |
| | | Phone: PPD |
| CRO Medical Monitor and | PPD | PPD |
| 24-Hour Emergency Contact | | PPD |
| | | 02-785 Warsaw, Poland |
| | | Mobile: PPD |
| | | Fax: PPD |
| SAE and Pregnancy Reporting | PPD Safety Medical Monitor | US Email: PPD |
| | | EU/Rest of World (ROW) Email: |
| | | PPD |
| | | US Fax Number: PPD |
| | | EU/ROW Fax Number: PPD |

Abbreviations: CRO=contract research organization; SAE=serious adverse event

Estimated date of last subject's last visit: O4 2018

## 2. SYNOPSIS

Name of Sponsor/Company: Alkermes, Inc.

Name of Investigational Product: ALKS 3831

Name of Active Ingredient: Olanzapine and samidorphan

Title of Study: A Phase 3, Multicenter Study to Assess the Long Term Safety and Tolerability of ALKS 3831 in Subjects with Schizophrenia

Investigators: This is a multinational, multicenter study.

Study Period:

Estimated date of first subject's consent: Q1 2016

#### **Objectives:**

**Primary:** The primary objective of this study is to evaluate the long-term safety and tolerability of ALKS 3831 in subjects with schizophrenia.

**Methodology:** Subjects that have completed the 4-week Treatment Period of the antecedent study, ALK3831-A305, within the past 7 days are eligible to be enrolled in this study. Subjects completing the antecedent study as inpatients may continue as inpatients for up to 1 week in this extension study. These subjects may be discharged from the inpatient unit at any time during this week based on Investigator's judgment.

Subjects enrolled in the study will be started on ALKS 3831 10/10 (10 mg olanzapine/10 mg samidorphan). The dose may be increased to ALKS 3831 15/10 (15 mg olanzapine/10 mg samidorphan) and up to ALKS 3831 20/10 (20 mg olanzapine/10 mg samidorphan) during the first week or thereafter, based on Investigator discretion. For subjects entering this study as outpatients, study staff will check in with them by phone on Day 3 to assess tolerability and determine if a dose increase is needed. An Unscheduled Visit will be arranged mid-Week 1 for subjects requiring a dose increase to ALKS 3831 15/10 or ALKS 3831 20/10. Following a dose increase, the dose may be decreased back to 10/10 or 15/10 if there are tolerability issues. Thus, dosing is flexible and subjects will receive ALKS 3831 10/10, 15/10, or 20/10 throughout the duration of the study, based on Investigator discretion. Dose adjustments can only be performed on-site at the study center. Subjects requiring dose adjustments between visits should arrange an Unscheduled Visit where the following procedures will be performed: study drug return, adherence review, and study drug dispensation.

Safety assessments will include adverse event (AE) monitoring, clinical laboratory testing, vital signs, weight and waist circumference assessments, 12-lead electrocardiograms (ECGs), movement disorder assessments, including the Abnormal Involuntary Movement Scale (AIMS), Barnes Akathisia Rating Scale (BARS), and Simpson Angus Scale (SAS), and the Columbia-Suicide Severity Rating Scale (C-SSRS).

Antipsychotic efficacy assessments to evaluate durability of treatment effect include Positive and Negative Syndrome Scale (PANSS) and Clinical Global Impressions-Severity (CGI-S).

Additional assessments include the Impact of Weight on Quality of Life-Lite Questionnaire (IWQOL-Lite), Cigarette Use, and EuroQOL-5D (EQ-5D).

Subjects completing 52 weeks of treatment with study drug will be eligible to continue in the open-label, long-term safety study (ALK3831-A308) and will continue to receive ALKS 3831. Subjects not continuing in the ALK3831-A308 long-term safety study will enter a 4-week Safety Follow-up Period. A schematic summarizing the study design is shown below.



\*Visits will occur weekly for the first 2 weeks, then biweekly thereafter. Outpatient subjects will be contacted by phone on Day 3 to determine if a dose increase is needed, and, if so, an unscheduled visit will be arranged mid-Week 1. The dose may be adjusted to either 10/10, 15/10, or 20/10 mg throughout the study period, based on Investigator discretion, and such dose adjustments will require subjects to visit the study site

**Number of Subjects Planned:** Approximately 390 subjects are planned to be enrolled in this study.

#### **Main Criteria for Inclusion:**

- 1. Subject is willing and able to provide informed consent; subject has signed the informed consent form before initiation of any study specific procedures
- 2. Subject agrees to use an acceptable method of contraception for the duration of the study
- 3. Subject is willing and able to follow the study procedures as outlined in the protocol
- 4. Subject has the potential to benefit from the administration of ALKS 3831, in the opinion of the Investigator
- 5. Subject has completed the antecedent study, ALK3831-A305, within 7 days

#### **Main Criteria for Exclusion:**

- 1. Subject has any finding that, in the view of the Investigator or Medical Monitor, would compromise the safety of the subject or affect their ability to fulfill the protocol visit schedule or visit requirement
- 2. Subject is currently taking medications that are contraindicated with olanzapine use or exhibit drug-interaction potential with olanzapine will be defined and prohibited at the discretion of the Principal Investigator (PI)
- 3. Subject has a positive test for drugs of abuse at study entry
- 4. Subject is pregnant, planning to become pregnant, or breastfeeding during the study

**Investigational Product, Dosage, Duration, and Mode of Administration:** ALKS 3831 will be supplied as a coated bilayer tablet containing either 10, 15, or 20 mg olanzapine and 10 mg samidorphan. The tablet is to be taken by mouth once daily, preferably at bedtime.

Reference Therapy, Dosage, Duration, and Mode of Administration: Not applicable.

**Duration of Study:** The study duration will be up to 56 weeks, which includes a 52-week Treatment Period and a 4-week Safety Follow-up Period.

#### **Criteria for Evaluation:**

#### Safety:

The safety assessments include:

- Adverse events (AEs)
- Clinical laboratory parameters (chemistry, hematology, and urinalysis)
- Vital signs (oral temperature, respiratory rate, orthostatic blood pressure, and pulse)
- Weight and waist circumference
- ECG parameters (heart rate, RR, PR, QRS, and QT)
- C-SSRS
- AIMS
- BARS
- SAS

#### **Efficacy:**

The efficacy assessments include:

- PANSS
- CGI-S

#### Other:

Other assessments include:

- IWQOL-Lite
- Cigarette Use
- EQ-5D

#### **Statistical Methods:**

The Safety Population is defined as all enrolled subjects who receive at least one dose of ALKS 3831 in this study. The Full Analysis Set (FAS) Population is defined as all subjects that receive at least one dose of ALKS 3831 and at least one postdose PANSS assessment in this study.

Safety analyses will be carried out using the Safety Population. Incidence of AEs will be analyzed as a safety endpoint. Reported AE terms will be coded using the Medical Dictionary for Regulatory Activities (MedDRA®) and will be summarized by system organ class and preferred term categories. Serious AEs and AEs leading to study discontinuation (AEDCs) will also be summarized.

Observed values and changes from Baseline in weight, body mass index (BMI), waist circumference, laboratory parameters, vital signs, and ECG parameters will be summarized by study visit. Prior and concomitant medication use will be summarized by World Health Organization (WHO) Drug Dictionary Anatomical Therapeutic Class (ATC) code.

Efficacy analyses will be carried out using the FAS Population. The following efficacy endpoints will be analyzed to evaluate the durability of treatment effect for ALKS 3831:

- Change from Baseline in PANSS total score and subscales by visit
- Change from Baseline in CGI-S by visit
- PANSS response
- Relapse
- Remission

#### • Time to discontinuation

The PANSS (total and subscale scores) and CGI-S scores, and appropriate changes from Baseline, will be summarized using descriptive statistics. Positive and Negative Syndrome Scale response and remission at each visit will be summarized as number and percentage.

The discontinuation rate and the relapse rate will be estimated using the Kaplan-Meier (KM) Method and the KM plot will be provided.

**Sample Size Considerations:** Approximately 390 subjects are planned to be enrolled in this study.

| <b>3.</b> | TABLE OF CONTENTS | |
|-----------|--------------------------------------|----|
| 1. | TITLE PAGE | 1 |
| 2. | SYNOPSIS | 3 |
| 3. | TABLE OF CONTENTS | 7 |
| 4. | LIST OF ABBREVIATIONS | 11 |
| 5. | INTRODUCTION | 13 |
| 5.1. | Background | 13 |
| 5.2. | Study Drugs | 14 |
| 5.2.1. | Samidorphan | 14 |
| 5.2.2. | Olanzapine | 14 |
| 5.3. | Study Rationale | 15 |
| 5.4. | Dose Rationale | 15 |
| 6. | OBJECTIVES | 16 |
| 6.1. | Primary Objective | 16 |
| 7. | SELECTION AND WITHDRAWAL OF SUBJECTS | 17 |
| 7.1. | Subject Inclusion Criteria | 17 |
| 7.2. | Subject Exclusion Criteria | 17 |
| 7.3. | Subject Withdrawal | 17 |
| 7.4. | Replacement of Subjects | 18 |
| 8. | STUDY DESIGN | 19 |
| 8.1. | Overall Study Design and Plan. | 19 |
| 8.2. | Schedule of Visits and Assessments | 20 |
| 8.3. | Study Procedures Descriptions | 24 |
| 8.3.1. | Informed Consent | 24 |
| 8.3.2. | Eligibility Review | 24 |
| 8.3.3. | Demographics and Medical History | 24 |
| 8.3.4. | Concomitant Medication Review | 24 |
| 8.3.5. | Vital Signs | 24 |
| 8.3.6. | Physical Examination | 25 |
| 8.3.7. | Body Weight and Waist Circumference | 25 |
| 8.3.8. | 12-Lead Electrocardiogram | 25 |

| 8.3.9. | Structured Interviews and Questionnaires | 25 |
|-----------|---------------------------------------------------------|----|
| 8.3.9.1. | Antipsychotic Efficacy Assessments | 25 |
| 8.3.9.2. | Safety Assessments | 26 |
| 8.3.9.3. | Other Assessments | 26 |
| 8.3.10. | Laboratory Assessments | 27 |
| 8.3.10.1. | Drug Testing | 27 |
| 8.3.10.2. | Hematology, Biochemistry, and Urinalysis | 27 |
| 8.3.10.3. | Pregnancy Testing | 28 |
| 8.3.11. | Drug Dispensation and Reconciliation | 29 |
| 8.3.12. | Emergency Treatment Card | 29 |
| 8.3.13. | Adverse Event Monitoring | 29 |
| 8.4. | Study Requirements and Restrictions | 29 |
| 8.4.1. | Contraception and Pregnancy | 29 |
| 8.4.2. | Prohibited Medications | 30 |
| 8.4.3. | Permitted Therapy | 31 |
| 8.4.4. | Pain Management | 31 |
| 8.4.5. | Other Restrictions and Requirements | 32 |
| 9. | TREATMENT OF SUBJECTS | 33 |
| 9.1. | Study Drug Dose and Administration | 33 |
| 9.2. | Treatment Adherence. | 33 |
| 9.3. | Randomization/Method of Assigning Subjects to Treatment | 33 |
| 9.4. | Blinding | 33 |
| 10. | STUDY DRUG MATERIALS AND MANAGEMENT | 34 |
| 10.1. | Study Drug | 34 |
| 10.2. | Packaging and Labeling | 34 |
| 10.3. | Storage | 34 |
| 10.4. | Accountability | 34 |
| 10.5. | Handling and Disposal | 35 |
| 11. | ASSESSMENT OF EFFICACY | 36 |
| 12. | ASSESSMENT OF PHARMACOKINETICS AND PHARMACODYNAMICS | 37 |
| 13. | ASSESSMENT OF SAFETY | 38 |
| 13.1. | Definition of Adverse Event | 38 |

| 13.2. | Definition of Serious Adverse Event | 38 |
|-----------|---------------------------------------------------------|----|
| 13.3. | Relationship to Study Drug | 39 |
| 13.4. | Monitoring and Recording of Adverse Events | |
| 13.5. | Reporting of Serious Adverse Events and Pregnancy | 41 |
| 14. | STATISTICS | 43 |
| 14.1. | Sample Size Considerations | 43 |
| 14.2. | General Statistical Methodology | 43 |
| 14.2.1. | Study Population | 43 |
| 14.2.1.1. | Safety Population | |
| 14.2.1.2. | Full Analysis Set | 43 |
| 14.3. | Demographics and Baseline Data | 43 |
| 14.4. | Safety and Tolerability Analyses | 43 |
| 14.5. | Efficacy Analysis | 44 |
| 14.6. | Pharmacokinetic/Pharmacodynamic Analyses | 44 |
| 15. | DIRECT ACCESS TO SOURCE DATA/DOCUMENTS | 45 |
| 15.1. | Study Monitoring | 45 |
| 15.2. | Audits and Inspections | 45 |
| 15.3. | Institutional Review Board/Independent Ethics Committee | 45 |
| 16. | QUALITY CONTROL AND QUALITY ASSURANCE | 46 |
| 16.1. | Case Report Forms | 46 |
| 16.2. | Confidentiality of Data | 46 |
| 17. | ETHICAL CONSIDERATIONS | 47 |
| 17.1. | Ethics Review | 47 |
| 17.2. | Ethical Conduct of the Study | 47 |
| 17.3. | Written Informed Consent | 47 |
| 18. | DATA HANDLING AND RECORDKEEPING | 49 |
| 18.1. | Data Capture | 49 |
| 18.2. | Inspection of Records | 49 |
| 18.3. | Retention of Records | 49 |
| 18.4. | Use of Information and Publication Policy | 50 |
| 19. | REFERENCES | 51 |
| 20. | APPENDICES | 53 |

# LIST OF TABLES

| Table 1: | Study Contact Information | 2 |
|---|---|---|
| Table 2: | List of Abbreviations and Definitions of Terms | 11 |
| Table 3: | Schedule of Assessments | 21 |
| Table 4: | Clinical Laboratory Assessments | 28 |
| Table 5: | Adverse Event Causality Guidelines | 40 |
| | LIST OF FIGURES | |
| Figure 1: | Study Design Schematic | 20 |
| | LIST OF APPENDICES | |
| Appendix A | Partial List of Prohibited Cytochrome P450 (CYP) 3A4 Inhibitors | and Inducers |
| Appendix B | Positive and Negative Syndrome Scale | |
| Appendix C | C: Clinical Global Impression | |
| | <ul> <li>Severity</li> </ul> | |
| Appendix D | Abnormal Involuntary Movement Scale | |
| Appendix E | Barnes Akathisia Rating Scale | |
| Appendix F | Simpson-Angus Scale | |
| Appendix C | G: Columbia-Suicide Severity Rating Scale | |
| | <ul> <li>Since Last Visit</li> </ul> | |
| Appendix H | I: Impact of Weight on Quality of Life-Lite | |
| Appendix I | : EuroQOL-5D | |

## 4. LIST OF ABBREVIATIONS

The following abbreviations are used in this study protocol.

**Table 2:** List of Abbreviations and Definitions of Terms

| Abbreviation or Term | Explanation or Definition |
|---|---|
| AE | Adverse event |
| AIMS | Abnormal Involuntary Movement Scale |
| ATC | Anatomical Therapeutic Chemical [classification system] |
| BARS | Barnes Akathisia Rating Scale |
| BMI | Body mass index |
| CGI-S | Clinical Global Impression-Severity |
| CRO | Contract research organization |
| CSA | Clinical Study Agreement |
| C-SSRS | Columbia-Suicide Severity Rating Scale |
| EC | Ethics Committee |
| ECG | Electrocardiogram |
| eCRF | Eectronic case report form |
| EOT | End of treatment |
| EQ-5D | EuroQOL-5D |
| ET | Early termination |
| FAS | Full analysis set |
| GCP | Good Clinical Practice |
| HbA1C | Hemoglobin A1c |
| ICF | Informed consent form |
| ICH | International Conference on Harmonisation of Technical Requirements for Registration of Pharmaceuticals for Human Use |
| IWQOL | Impact of Weight on Quality of Life |
| IRB | Institutional Review Board |
| KM | Kaplan-Meier |
| MedDRA | Medical Dictionary for Regulatory Activities |
| PANSS | Positive and Negative Syndrome Scale |
| PCP | Phencyclidine |
| PI | Principal Investigator |
| SAE | Serious adverse event |
| SAS | Simpson-Angus Scale |

# Table 2: List of Abbreviations and Definitions of Terms (Continued)

| Abbreviation or Term | Explanation or Definition |
|----------------------|---------------------------|
| WHO | World Health Organization |

## 5. INTRODUCTION

## 5.1. Background

Schizophrenia is a chronic, severe disease with debilitating psychotic symptoms, physical and psychiatric comorbidities, and increased mortality. Despite the availability of a range of FDA-approved medicines, the disease is still inadequately treated, and is associated with enormous human and economic cost. Life expectancy is reduced by 19 years in men and 16 years in women with schizophrenia compared to the general population (Harris and Barraclough 1998; Lambert et al, 2010; Tiihonen et al, 2009). The decreased life expectancy is due to a combination of direct effects of the disease, eg, increased rates of suicide and violence (Hodgins 2008; Kuo et al, 2005), as well as indirect causes, including increased incidence of obesity and cardiovascular disease (Nasrallah et al, 2006; Saha et al, 2007).

The goal of treatment in schizophrenia is to achieve the maximal reduction in positive and negative symptoms and increase functionality. Unfortunately, even with regular administration of currently available antipsychotic medications at full therapeutic dose levels, the overwhelming majority of patients continue to exhibit residual active symptomatology. For physicians and patients, in many cases the current treatment paradigm involves an efficacy/tolerability trade-off, where use of the most efficacious agents is avoided or delayed in order to avoid known safety issues. As such, there is a need for more efficacious therapies with better tolerability.

Olanzapine is regarded as one of the most effective antipsychotic agents with well-recognized efficacy and decreased incidence of extrapyramidal symptoms. However, its efficacy is compromised by safety and tolerability limitations that affect compliance and retention of patients on olanzapine therapy (Lieberman et al, 2005). In particular, results of the Clinical Antipsychotic Trials of Intervention Effectiveness (CATIE), identify olanzapine as an effective atypical antipsychotic associated with the highest weight gain (9.4 kg increase over a treatment period up to 18 months and  $\geq$ 7% body weight in 30% of subjects) and a comparatively higher discontinuation rate relative to other antipsychotic agents due to weight gain and metabolic effects. As a result of these limitations surrounding safety, tolerability, adherence, and retention, the risk of olanzapine therapy can outweigh the benefit, and patients are often switched to alternative antipsychotic agents even if they are less effective.

ALKS 3831 is a fixed-dose combination product of olanzapine and samidorphan (a μ-opioid antagonist) under investigation for the treatment of schizophrenia. Phase 1 and Phase 2 studies demonstrated that coadministration of samidorphan with olanzapine attenuates the weight gain experienced with olanzapine alone. Results from these studies are described in more detail in Section 5.3. ALKS 3831 may have the further benefit of controlling substance abuse in patients with schizophrenia. Comorbid substance use disorder is a well-recognized obstacle to patient care. An estimated 1 out of every 3 patients with schizophrenia (33.7%) meet or have met criteria for alcohol use disorder (Regier et al, 1990). Patients with both schizophrenia and alcohol use disorder represent a common variant within the schizophrenia spectrum that is difficult to treat and is associated with an extremely poor prognosis (Dixon 1999; Koekkoek et al, 2006). Samidorphan (also referred to as ALKS 33 or RDC-0313), is structurally derived from naltrexone and is a potent μ-opioid antagonist. In clinical studies, it has been shown to block

both the subjective and physiological effects of the opioid agonist remifentanil (ALK33-004) and it is correlated with reduced drinking behavior in adults with alcohol dependence (ALK33-005). ALK3831-401 is an ongoing clinical study designed to evaluate the effect of ALKS 3831 on drinking behavior in adult subjects with schizophrenia and alcohol use disorder.

In summary, ALKS 3831 is being explored as a therapeutic agent for the treatment of schizophrenia designed to combine the antipsychotic efficacy of olanzapine with a reduced risk of weight gain and associated metabolic deficits. Development of ALKS 3831 as a fixed-dose combination of olanzapine and samidorphan has the potential to improve upon the benefit/risk profile of olanzapine alone and address a significant clinical need for patients that are currently forced to choose between treatment efficacy and safety.

## 5.2. Study Drugs

In this study, a fixed-dose combination of olanzapine and samidorphan will be administered in a single bilayer tablet. The following sections provide an overview of samidorphan and olanzapine. Detailed information about the study drugs can be found in the current ALKS 3831 Investigator's Brochure.

## 5.2.1. Samidorphan

Samidorphan is a new chemical entity in clinical development by Alkermes. It is an opioid modulator which acts primarily as an antagonist at  $\mu$  opioid receptors, with mixed agonist/antagonist activity at  $\delta$  and  $\kappa$  receptors. It is currently being investigated in combination with buprenorphine for the treatment of major depressive disorder (ALKS 5461) and in combination with olanzapine for the treatment of schizophrenia. Based on its chemical structure, samidorphan is considered a Schedule II controlled substance according to the US Drug Enforcement Agency and will require proper handling (see Section 10). At least ten clinical studies of samidorphan have been conducted to date, eight of which included subjects that received samidorphan alone (not in combination with another product). Commonly reported adverse events (AEs) observed across all studies included nausea, fatigue, and somnolence. Overall, no trends or clinically meaningful changes have been observed in clinical laboratory analytes, vital sign parameters, or electrocardiogram (ECG) data.

## 5.2.2. Olanzapine

Olanzapine has been available in the US since 1996 (Zyprexa®) and was originally approved for the treatment of schizophrenia. It has since been approved for other indications, including the treatment of schizophrenia in adolescents and bipolar disorder. The safety and tolerability profile of olanzapine is well documented, and AE labeling is supported by an extensive safety database that includes over 8,500 adult patients (Eli Lilly and Company 2017). Commonly reported AEs consistent across all or most dosage forms in short-term, placebo controlled trials include somnolence, constipation, dry mouth, accidental injury, weight gain, postural hypotension, dizziness, asthenia, fever, and abnormal gait.

## **5.3.** Study Rationale

Phase 1 and Phase 2 studies (ALK33-301 and ALK3831-302, respectively) have demonstrated that ALKS 3831 significantly attenuates olanzapine-induced weight gain while providing similar antipsychotic efficacy for stabilization of schizophrenia symptoms. Safety and tolerability data from these studies indicate that ALKS 3831 is safe and generally well-tolerated. However, the longest treatment period assessed to date is 24 weeks. The proposed study will extend these findings and evaluate the safety and tolerability of ALKS 3831 over a 52-week period.

#### **5.4.** Dose Rationale

The selected doses of ALKS 3831 (10/10 [10 mg olanzapine/10 mg samidorphan], 15/10 [15 mg olanzapine/10 mg samidorphan], and 20/10 [20 mg olanzapine/10 mg samidorphan]) are within the approved olanzapine therapeutic dose range for the treatment of schizophrenia (Eli Lilly and Company 2017) and represent the intended commercial doses of ALKS 3831.

The 10 mg samidorphan dose was identified as the minimally effective dose based on the robust efficacy and optimal safety profile observed in a previous Phase 2 study (ALK3831-302) with that dose. A fixed dose of samidorphan was selected due to the fact that data from this study demonstrated no correlation between the ratio of samidorphan/olanzapine dose and percent change from Baseline in body weight, indicating that even with higher olanzapine doses, a fixed dose of samidorphan is sufficient to achieve maximal effect on reducing olanzapine-induced weight gain.

# 6. **OBJECTIVES**

# 6.1. Primary Objective

The primary objective of this study is to evaluate the long-term safety and tolerability of ALKS 3831 in subjects with schizophrenia.

#### 7. SELECTION AND WITHDRAWAL OF SUBJECTS

## 7.1. Subject Inclusion Criteria

Each subject must meet all of the following inclusion criteria to be qualified to participate in this study.

- 1. Subject is willing and able to provide informed consent; subject has signed the informed consent form before initiation of any study specific procedures
- 2. Subject agrees to use an acceptable method of contraception for the duration of the study (please refer to Section 8.4.1 for additional details regarding contraception)
- 3. Subject is willing and able to follow the study procedures as outlined in the protocol
- 4. Subject has the potential to benefit from the administration of ALKS 3831, in the opinion of the Investigator
- 5. Subject has completed the 4-week Treatment Period (all visits up to and including Visit 6, End of Treatment) in the antecedent study, ALK3831-A305, within 7 days

## 7.2. Subject Exclusion Criteria

Each subject must not have any of the following conditions to be qualified to participate in this study.

- 1. Subject has any finding that, in the view of the Investigator or Medical Monitor, would compromise the safety of the subject or affect their ability to fulfill the protocol visit schedule or visit requirement
- 2. Subject is currently taking medications that are contraindicated with olanzapine use or exhibit drug-interaction potential with olanzapine will be defined and prohibited at the discretion of the Principal Investigator (PI)
- 3. Subject has a positive test for drugs of abuse at study entry
- 4. Subject is pregnant, planning to become pregnant, or breastfeeding during the study

## 7.3. Subject Withdrawal

A subject may be discontinued from the study at any time if the subject, Investigator, or the Sponsor determines that it is not in the best interest of the subject to continue participation. If a subject has an absolute neutrophil count (ANC)  $<1.0\times10^3$  per  $\mu$ L or HbA1c  $\ge6.5\%$  at any time during this extension study, the subject will be discontinued from the study. Other reasons for discontinuation include the following:

- AEs
- Lack of Efficacy
- Lost to follow-up
- Withdrawal by subject

- Protocol Deviation (noncompliance with study drug or study procedures)
- Pregnancy
- Study terminated by Sponsor
- Other

If a subject withdraws from the study for any reason, any ongoing AEs will be followed until resolution, until deemed stable by the Investigator, or until the subject is deemed by the Investigator to be lost to follow-up. If, in the opinion of the Investigator, it is necessary to monitor a subject beyond the Safety Follow-up Visit, the Follow-up Period may be extended, as necessary. In such instances, the Sponsor and the Investigator will agree to an acceptable follow-up schedule.

In the event that a subject chooses to withdraw from the study, the Investigator should make a reasonable effort to ascertain the reason(s) for withdrawal, while fully respecting the subject's rights. Enrolled subjects are to be asked to return to the clinic for an Early Termination (ET) Visit and to complete a subsequent Safety Follow-up Period. The ET Visit should be scheduled as close as possible to the subject's last dose and will mimic the assessments scheduled to be conducted at the End of Treatment (EOT) Visit (Visit 28, Table 3). If the subject fails or refuses to return to the study center, an attempt must be made to contact the subject by telephone in order to assess as many safety and efficacy parameters as possible. All data collected over the telephone must be documented and kept in the subject's record.

The Investigator must maintain a record of all subjects who fail to complete the study. The reason for study discontinuation will be documented and entered on the appropriate electronic case report form (eCRF). If a subject is lost to follow-up, a reasonable attempt to contact the subject must be made and documented.

## 7.4. Replacement of Subjects

Subjects prematurely discontinued from the study will not be replaced.

#### 8. STUDY DESIGN

## 8.1. Overall Study Design and Plan

Subjects that have completed the 4-week Treatment Period of the antecedent study, ALK3831-A305, within the past 7 days are eligible to be enrolled in the study. Subjects completing the 4-week Treatment Period of the antecedent study, ALK3831-A305, as inpatients may continue as inpatients for up to 1 week in this extension study. These subjects may be discharged from the inpatient unit at any time during this week based on Investigator's judgment.

Subjects enrolled in the study will be started on ALKS 3831 10/10 (10 mg olanzapine/10 mg samidorphan). The ALKS 3831 dose may be increased to 15/10 (15 mg olanzapine/10 mg samidorphan) or 20/10 (20 mg olanzapine/10 mg samidorphan) during the first week of treatment or thereafter, based on Investigator discretion. For subjects entering this study as outpatients, study staff will check in with them by phone on Day 3 to assess tolerability and determine if a dose increase to ALKS 3831 15/10 or 20/10 is needed. An Unscheduled Visit will be arranged mid-Week 1 for subjects requiring a dose increase. Following a dose increase, the dose may be decreased back to 15/10 or 10/10 if there are tolerability issues. Thus, dosing is flexible and subjects will receive ALKS 3831 10/10, 15/10, or 20/10 throughout the duration of the study, based on Investigator discretion. Dose adjustments can only be performed on-site at the study center. Subjects requiring dose adjustments between scheduled visits should arrange an Unscheduled Visit for the following procedures: study drug return, adherence review, and study drug dispensation.

Safety assessments will include AE monitoring, clinical laboratory testing, vital signs, weight and waist circumference assessments, 12-lead ECGs, movement disorder assessments, including the Abnormal Involuntary Movement Scale (AIMS), Barnes Akathisia Rating Scale (BARS), and Simpson Angus Scale (SAS), and the Columbia-Suicide Severity Rating Scale (C-SSRS).

Efficacy assessments to evaluate the durability of treatment effect will include Positive and Negative Syndrome Scale (PANSS) and Clinical Global Impressions-Severity (CGI-S).

Additional assessments include Impact of Weight on Quality of Life–Lite Questionnaire (IWQOL-Lite), Cigarette Use, and EuroQOL-5D (EQ-5D).

Subjects completing 52 weeks of treatment with study drug will be eligible to continue in the open-label, long-term safety study (ALK3831-A308) and will continue to receive ALKS 3831. Subjects not continuing in the ALK3831-A308 long-term safety study will enter a 4-week Safety Follow-up Period. The overall schedule of visits and assessments for each Treatment Group is provided in Table 3.

A schematic of the study design is provided in Figure 1.

Figure 1: Study Design Schematic



\*Visits will occur weekly for the first 2 weeks, then biweekly thereafter. Outpatient subjects will be contacted by phone on Day 3 to determine if a dose increase is needed, and, if so, an unscheduled visit will be arranged mid-Week 1. The dose may be adjusted to either 10/10, 15/10, or 20/10 mg throughout the study period, based on Investigator discretion, and such dose adjustments will require subjects to visit the study site

## 8.2. Schedule of Visits and Assessments

The schedule of assessments is shown in Table 3.

A visit window of  $\pm 2$  days is permitted throughout the Treatment Period and the Follow-up Period (Visits 2-30). For a missed visit, the site should attempt to contact the subject to reschedule.

Premature discontinuation procedures are provided in Section 7.3.

On Day 3, study staff will check in with outpatient subjects by phone to determine if a dose increase to ALKS 3831 15/10 or 20/10 is needed. If, in the opinion of the Investigator, a dose increase is warranted, an Unscheduled Visit will be arranged mid-Week 1. The following procedures will be performed during the Unscheduled Visit: study drug return, adherence review, and study drug dispensation.

Dose adjustments can only occur on-site and require subjects to come to the study center. Throughout the study, subjects requiring dose adjustments between scheduled visits may arrange an Unscheduled Visit (same procedures as mid-Week 1 Unscheduled Visit described above).

**Table 3:** Schedule of Assessments

| | | | | | | | | | | | | 0 | pen l | Label | Trea | tmen | t Peri | od | | | | | | | | | | | u | low-<br>ip<br>riod |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Visit <sup>a</sup> | <b>1</b> <sup>b</sup> | <b>2</b> ° | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | 13 | 14 | 15 | 16 | 17 | 18 | 19 | 20 | 21 | 22 | 23 | 24 | 25 | 26 | 27 | 28/<br>ET/<br>EOT | 29 <sup>d</sup> | 30 |
| Study week | - | 1 | 2 | 4 | 6 | 8 | 10 | 12 | 14 | 16 | 18 | 20 | 22 | 24 | 26 | 28 | 30 | 32 | 34 | 36 | 38 | 40 | 42 | 44 | 46 | 48 | 50 | 52 | 54 | 56 |
| Informed<br>Consent | X | | | | | | | | | | | | | | | | | | | | | | | | | | | | | |
| Eligibility<br>Criteria | X | | | | | | | | | | | | | | | | | | | | | | | | | | | | | |
| Pregnancy<br>Testing <sup>e</sup> | X | | | | | | | X | | | | | | X | | | | | | X | | | | | | | | | | |
| Urine Drug<br>Screen | X | | | | | | | | | | | | | | | | | | | | | | | | | | | | | |
| Weight | | X | X | X | X | X | | X | | X | | X | | X | | X | | X | | X | | X | | X | | X | | X | | X |
| Waist<br>Circum-<br>ference | | X | X | X | X | X | | X | | X | | X | | X | | X | | X | | X | | X | | X | | X | | X | | X |
| Vital<br>Signs <sup>g</sup> | | X | X | X | X | X | | X | | X | | X | | X | | X | | X | | X | | X | | X | | X | | X | | X |
| Laboratory<br>Samples | | | | X | | | | X | | | | | | X | | | | | | X | | | | | | | | X | | |
| ECG | | | | X | | | | X | | | | | | X | | | | | | X | | | | | | | | X | | |
| Physical<br>Exam | | | | X | | | | X | | | | | | Х | | | | | | X | | | | | | | | X | | |
| PANSS <sup>i</sup> | | | | X | | X | | X | | | | | | X | | | | | | X | | | | | | | | X | | |
| CGI-S | | | | X | | X | | X | | X | | X | | X | | X | | X | | X | | X | | X | | X | | X | | |
| AE <sup>j</sup> | | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| ConMed <sup>j</sup> | | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| C-SSRS <sup>k</sup> | | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |

**Table 3:** Schedule of Assessments (Continued)

| | | | | | | | | | | | | Op | en La | ıbel T | reat | ment | Perio | d | | | | | | | | | | | - | low-<br>ip<br>riod |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Visit <sup>a</sup> | 1 <sup>b</sup> | 2° | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | 13 | 14 | 15 | 16 | 17 | 18 | 19 | 20 | 21 | 22 | 23 | 24 | 25 | 26 | 27 | 28/<br>ET/<br>EOT | <b>29</b> <sup>d</sup> | 30 |
| Study week | - | 1 | 2 | 4 | 6 | 8 | 10 | 12 | 14 | 16 | 18 | 20 | 22 | 24 | 26 | 28 | 30 | 32 | 34 | 36 | 38 | 40 | 42 | 44 | 46 | 48 | 50 | 52 | 54 | 56 |
| Abnormal<br>Movement<br>Scales | | | | X | | | | X | | | | | | X | | | | | | X | | | | | | | | X | | |
| IWQOL | X | | | X | | | | X | | | | | | X | | | | | | X | | | | | | | | X | | |
| EQ-5D | X | | | X | | | | X | | | | | | X | | | | | | X | | | | | | | | X | | |
| Cigarette<br>Use | X | | | X | | | | X | | | | | | X | | | | | | X | | | | | | | | X | | |
| Emergency<br>Treatment<br>Card <sup>m</sup> | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | | |
| Study Drug<br>Dispensation | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | | | |
| Study Drug<br>Adherence<br>Review | | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | D. ( | |

Abbreviations: AE=adverse event; CGI-S=Clinical Global Impression-Severity; ConMed=concomitant medication; C-SSRS=Columbia-Suicide Severity Rating Scale; ECG=electrocardiogram; EOT=End of Treatment; EQ-5D=EuroQOL-5D; IWQOL=Impact of Weight on Quality of Life; PANSS=Positive and Negative Syndrome Scale

<sup>&</sup>lt;sup>a</sup> A visit window of ±2 days is permitted throughout the Treatment Period and the Follow-up Period (Visits 2-30)

b Visit 1 must occur within 7 days of the EOT Visit (Visit 6) of the antecedent study, ALK3831-A305, and may occur on the same day. Assessments from ALK3831-A305 Visit 6 will constitute the Baseline/Screening assessments for this extension study

<sup>&</sup>lt;sup>c</sup> On Day 3, study staff will contact outpatient subjects by phone to determine if a dose increase to ALKS 3831 15/10 or 20/10 is needed. An Unscheduled Interim Visit will be arranged for subjects requiring a dose adjustment for study drug return and adherence review and study drug dispensation. Any subsequent dose adjustments throughout the study require subjects to come to the site for either a scheduled or unscheduled visit

<sup>&</sup>lt;sup>d</sup> Follow-up Visits (Visits 29 and 30) are not required for subjects who enroll in ALK3831-A308

<sup>&</sup>lt;sup>e</sup> Urine pregnancy test prior to dosing at Visit 1 and at all subsequent specified visits

- f Urine drug screen via dipstick prior to dosing on Day 1 for subjects who did not receive a urine drug screen at Visit 6 of the ALK3831-A305 study, or for subjects for whom Visit 1 of this study is not the same day as Visit 6 of the ALK3831-A305 study. Urine drug screen includes opiates, phencyclidine (PCP), amphetamine/methamphetamine, and cocaine
- g Vital signs include orthostatic blood pressure and heart rate, respiratory rate, and oral body temperature. Blood pressure, pulse rate, and respiratory rate will be taken after the subject has been supine for 5 minutes and once again after the subject has stood for 2 minutes
- h Subjects must fast (no food or drink except water) for at least 8 hours before laboratory draws. Laboratory draws are to be conducted in the morning for all specified visits
- <sup>1</sup> PANSS should be administered before other psychiatric assessments at each specified study visit
- <sup>j</sup> AEs ongoing at the end of the antecedent study or concomitant medications continuing from the antecedent study will be carried over and followed through until resolution
- <sup>k</sup> The "Since Last Visit" version to be used at all visits
- <sup>1</sup> Abnormal movement scales include the following: Abnormal Involuntary Movement Scale (AIMS), Barnes Akathisia Rating Scale (BARS), and Simpson-Angus Scale (SAS)
- <sup>m</sup> Emergency treatment card to be dispensed at Visit 1, confirmed at subsequent timepoints, and collected at Visit 28, EOT
- <sup>n</sup> Calls should be made in weeks between in-person study visits to ensure subjects are continuing to stay adherent with medication. An Unscheduled Visit will be arranged for any dose adjustments required between planned visits when subjects will come to the site for study drug return and new drug dispensation

## 8.3. Study Procedures Descriptions

Details of the study procedures are described below. The overall schedule of assessments is provided in Table 3. Information collected with the following assessments will be carried forward from the antecedent study, ALK3831-A305, for Screening/Baseline: demographics and medical history, vital signs, physical exam, height, body weight and waist circumference, 12-lead ECG, CGI-S, PANSS, and Abnormal Movement Scales.

#### 8.3.1. Informed Consent

The nature of the study and its risks and benefits will be explained to the subject by the Investigator or designated study personnel as outlined in Section 17.3.

Prior to the administration of any study-specific procedures, authorized study personnel will obtain written informed consent from each potential subject.

## 8.3.2. Eligibility Review

An eligibility review will be conducted by the Investigator at the visit specified in Table 3 using the subject inclusion criteria in Section 7.1 and exclusion criteria in Section 7.2.

## 8.3.3. Demographics and Medical History

Subjects' demographic data and medical history will be carried over from the antecedent study, ALK3831-A305.

#### **8.3.4.** Concomitant Medication Review

At the timepoints specified in Table 3, subjects will be asked about the medications they have taken since their last visit, including prescription and nonprescription medications, vitamins, and supplements.

The Investigator will record the following data on all medications used by the subject: name, dose, regimen, route of administration, start and stop dates, and the indication for use.

#### 8.3.5. Vital Signs

Vital signs (ie, blood pressure, heart rate, respiratory rate, and oral body temperature) will be assessed at the timepoints specified in Table 3. An effort will be made to consistently use the same arm (preferably the subject's dominant arm) to measure blood pressure and heart rate throughout the study. The blood pressure cuff will be calibrated per study site standard operating procedures (SOP). Automated measurement is preferred, but if performed manually, heart rate will be measured in the brachial artery for at least 30 seconds. Orthostatic blood pressure and heart rate will be collected in the following manner:

- Allow subject to be in a supine position for at least 5 minutes
- Measure blood pressure and heart rate
- Have subject stand for 2 minutes
- Measure blood pressure and heart rate

Vital signs may be collected at any time during a scheduled visit, unless otherwise noted.

### 8.3.6. Physical Examination

A physical examination will be performed at the timepoints specified in Table 3.

#### 8.3.7. Body Weight and Waist Circumference

Body weight and waist circumference will be measured at all the timepoints specified in Table 3.

For weight measurements, subjects should be asked to void immediately prior to measurement and should be dressed in a hospital gown with consistent under-attire for each measurement. Subjects should remove all personal items, such as watches and jewelry, and they should be weighed on the same scale for each measurement under the same conditions.

Both weight and waist circumference will be measured three consecutive times at each assessment and all measurements will be recorded in the eCRF

## 8.3.8. 12-Lead Electrocardiogram

A 12-lead ECG will be conducted at the timepoints specified in Table 3. All scheduled ECGs must be performed after the subject has rested quietly for at least 5 minutes in the supine position.

A qualified clinician will conduct ECGs and assess ECG results using equipment that has been calibrated according to the site's SOP. The following ECG parameters will be collected: pulse, RR, PR, QRS, QT, QT interval corrected using the Fridericia formula (QTcF), and QT interval corrected using the Bazett formula (QTcB).

Electrocardiograms will also be evaluated by a central reader.

#### 8.3.9. Structured Interviews and Questionnaires

Brief descriptions of each of the interviews and questionnaires to be distributed are available below. All interviews and questionnaires will be administered by trained and qualified study personnel.

For assessments performed at multiple visits, every effort should be made to pair the same clinician/rater with the same subject across visits.

Table 3 provides information on the timepoints at which each assessment should be administered. For all visits where assessments overlap, the PANSS should be administered first before any other psychiatric assessment.

#### 8.3.9.1. Antipsychotic Efficacy Assessments

#### 8.3.9.1.1. Positive and Negative Syndrome Scale

The PI or designee will complete the PANSS (Appendix B) (Kay et al, 1987) according to the schedule in Table 3. The Structured Clinical Interview for the PANSS (SCI-PANSS) will be used to administer the PANSS.

### 8.3.9.1.2. Clinical Global Impression-Severity

The PI or designee will complete the CGI-Severity (CGI-S, Appendix C) scale at the timepoints specified in Table 3. The CGI-S measures mental illness severity. Clinicians are asked to rate subjects based on their prior experience working with individuals in a similar patient population (Guy 1976).

#### 8.3.9.2. Safety Assessments

#### 8.3.9.2.1. Abnormal Movement Rating Scales

The PI or designee will complete the following abnormal movement rating scales: The AIMS (Appendix D) (Guy 1976), the BARS (Appendix E) (Barnes 1989), and the SAS (Appendix F) (Simpson and Angus 1970) at the timepoints specified in Table 3.

After administration of the first dose of study drug, if a subject complains of extrapyramidal symptoms on a day when abnormal movement scale assessments are not scheduled, an unscheduled abnormal movement assessment should be performed.

## 8.3.9.2.2. Columbia-Suicide Severity Rating Scale

The PI or designee will administer the C-SSRS (Appendix G) according to the schedule in Table 3. The "Since Last Visit" version is to be completed at all scheduled timepoints. The C-SSRS should be administered by a qualified clinician trained in assessing and managing suicidal ideation and behavior (Posner et al, 2011).

#### 8.3.9.3. Other Assessments

#### **8.3.9.3.1.** Cigarette Use

Data on cigarette use will be collected using the question: "How many packs of cigarettes did you smoke over the past 7 days?" at the timepoints specified in Table 3.

#### 8.3.9.3.2. Impact of Weight on Quality of Life-Lite

Subjects will complete the IWQOL-Lite questionnaire (Appendix H) at the timepoints specified in Table 3.

#### 8.3.9.3.3. EuroQOL-5D

Subjects will complete the EQ-5D (Appendix I) at the timepoints specified in Table 3. This scale provides an indication of health status based on self-rating in the following five categories: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Additionally, it asks subjects to rank their health status on a visual analogue scale (VAS) from "worst imaginable health state" to "best imaginable health state."

## **8.3.10.** Laboratory Assessments

## **8.3.10.1. Drug Testing**

A drug screen for opiates (including codeine, hydrocodone, hydromorphone, methadone, morphine, oxycodone, and oxymorphone) and drugs of abuse (including amphetamine/methamphetamine, phencyclidine [PCP], and cocaine) will be performed at the timepoints specified in Table 3. Urine drug screens may be repeated based on Investigator judgment. The test may also be repeated at any time during the study, should the Investigator feel it is warranted. Subjects are not eligible for participation if the results are positive at Screening. If a subject is determined to be using any of these substances during the Treatment Period, the Investigator should contact the Medical Monitor to discuss the course of action.

## 8.3.10.2. Hematology, Biochemistry, and Urinalysis

Fasting blood and urine samples will be collected at the timepoints specified in Table 3 for specific hematology, biochemistry, and urinalysis assessments listed in Table 4. Subjects will be instructed not to eat or drink anything (except water) for 8 hours before each visit where blood samples for biochemistry and hematology assessments will be collected. Samples will be collected in accordance with the site's standard procedures and analyzed by a central laboratory. Laboratory assessments may be repeated at the Investigator's discretion.

**Table 4: Clinical Laboratory Assessments** 

| Hematology | Biochemistry | Urinalysis |
|---|---|---|
| Hematocrit | <b>General Chemistry</b> | Bilirubin |
| Hemoglobin | Albumin | Color and appearance |
| Platelet count | Bicarbonate | Glucose |
| Red blood cell count | Calcium | Ketones |
| Total and differential | Chloride | Leukocytes |
| (absolute) white blood cell | Creatine phosphokinase | Nitrite |
| count | Glucose | Occult blood |
| | Lactic dehydrogenase | pН |
| | Potassium | Protein |
| | Sodium | Specific gravity |
| | Total protein | Urobilinogen |
| | Uric acid | Cotinine |
| | <b>Endocrine Function Test</b> | |
| | HbA1c | Microscopic examination of |
| | Prolactin | sediment, only if urinalysis |
| | Insulin | dipstick results are abnormal |
| | <b>Liver Function Tests</b> | |
| | Alanine aminotransferase | |
| | Alkaline phosphatase | |
| | Aspartate aminotransferase | |
| | Gamma-glutamyl transferase | |
| | Total bilirubin | |
| | <b>Renal Function Tests</b> | |
| | Blood urea nitrogen | |
| | Creatinine | |
| | Lipid Panel | |
| | High-density lipoprotein | |
| | Low-density lipoprotein | |
| | Total cholesterol | |
| | Triglycerides | |

## 8.3.10.3. Pregnancy Testing

A urine pregnancy test will be administered to all women at the timepoints specified in Table 3. At Visit 1, results must be negative for the subject to be eligible for the study. As highlighted in Section 7.3 a positive pregnancy test result at any time will necessitate the subject's immediate withdrawal from the study. Additional follow-up may be necessary as indicated in Section 8.4.1.

## 8.3.11. Drug Dispensation and Reconciliation

Section 9 provides information related to drug dispensing procedures. Study drug will be dispensed/administered at the timepoints specified in Table 3. The study drug use and storage information will be explained to/reviewed with the subject.

Whether or not samidorphan is classified as a controlled substance varies from country to country; some countries have classified samidorphan as a controlled substance, while others have not. Sites will be given storage, handling, and reconciliation instructions applicable to their country to ensure compliance with local regulations for controlled substances.

## **8.3.12.** Emergency Treatment Card

An emergency treatment card will be distributed to each subject and collected from each subject at the timepoints indicated in Table 3. The card will indicate that the subject is receiving an opioid antagonist and olanzapine, and will include the PI's contact information, a suggested pain management plan and information regarding opiate blockade. Subjects will be instructed to keep the card with them at all times. Study personnel will confirm that subjects have the card in their possession at each study visit, as indicated in Table 3.

### **8.3.13.** Adverse Event Monitoring

Adverse events will be monitored continuously from the time a subject signs the informed consent document until the completion of the final study visit (see Table 3). Adverse events and serious AEs (SAEs) are defined in Section 13.1 and 13.2, respectively. Section 13.4 provides guidance on the monitoring and recording requirements for AEs. Section 13.5 provides guidance on the reporting requirements for SAEs.

## 8.4. Study Requirements and Restrictions

#### **8.4.1.** Contraception and Pregnancy

All male and female subjects must agree to use an acceptable method of contraception for the duration of the study unless they are surgically sterile or postmenopausal (see below). The following are considered acceptable methods of contraception:

- 1. Double-barrier protection (eg, a condom with spermicide or a diaphragm with spermicide)
- 2. Intrauterine device (IUD)
- 3. Oral contraceptive pills and other hormonal methods (eg, a vaginal ring, contraceptive patch, contraceptive implant); oral contraceptives should be initiated at least 30 days prior to Screening

Subjects who are abstinent are eligible, provided they agree to use an acceptable contraceptive method should they become sexually active.

Subjects who are surgically sterile are exempt from the requirement to use contraception. Women who have undergone a hysterectomy, bilateral tubal ligation, or bilateral salpingo-oophorectomy are considered surgically sterile. Men who have undergone a vasectomy

are considered surgically sterile. Partner vasectomy is not considered an approved acceptable method of contraception for a female subject.

Women who are postmenopausal are also exempt from the requirement to use contraception. For the purpose of this study, postmenopausal is defined as the permanent cessation of menstruation for at least 12 months prior to Screening in women who are 45 years of age or older.

If a subject becomes pregnant while participating in the study, she will be discontinued from study drug immediately. Additional follow-up may be required. Pregnancies in female subjects and female partners of male subjects should also be reported and will be followed in the same manner. A Pregnancy Report Form must be submitted to Alkermes via PPD (fax number in Section 13.5) immediately, within 24 hours of awareness of the pregnancy, irrespective of whether an AE has occurred. The pregnancy will be followed until completion or termination. If the outcome of the pregnancy meets the criteria for classification as a SAE it should be reported following the SAE procedure (see Section 13.5).

#### **8.4.2.** Prohibited Medications

The prohibited medications include the following:

- Monoamine oxidase inhibitors (eg, phenelzine, tranylcypromine, selegiline, or moclobemide)
- Long-acting formulations of any antipsychotic agent
- Use of antipsychotic sleep aids (eg, Seroquel) is prohibited. However, use of benzodiazepines to treat some symptoms is permissible
- In general, the use of psychotropic medications other than study drug is prohibited, with the exception of the following (these medications should only be administered after all assessments have been completed for that visit):
  - Beta-blockers (eg, propranolol or pinodolol), antihistamines, and anticholinergics may be used for treatment-emergent akathisia
  - Anticholinergies may be used for extrapyramidal symptoms
- Chantix<sup>®</sup> (varenicline) is not permitted. However, nicotine replacement therapy, including nicotine replacement patch and oral nicotine gum, is permitted
- All prescription or over-the-counter (OTC) agents taken for the purpose of weight reduction
- Systemic steroids administered by oral, intravenous, or intramuscular route
- Topiramate (Topamax<sup>®</sup>) and combination products containing topiramate; calcitonin (eg, Miacalcin<sup>®</sup>)
- Diabetes treatments and hypoglycemic agents including Metformin and Insulin

Medications that are contraindicated with olanzapine use or exhibit drug-interaction potential with olanzapine are prohibited.

Use of moderate-to-strong inhibitors or inducers of cytochrome P450 (CYP) 3A4 (prescription medications, OTC medications, or dietary supplements) is prohibited in the antecedent study and

is prohibited in this study throughout the Treatment Period and throughout Follow-up. Refer to Appendix A for a list of CYP3A4 inhibitors and inducers (Food and Drug Administration 2016; University of Washington: School of Pharmacy 2017a; University of Washington: School of Pharmacy 2017b).

The contract research organization (CRO) Medical Monitor should be consulted for any questions about use of any psychotropic medications during a subject's participation in this study.

Use of opioid antagonists, including naltrexone (any formulations) and naloxone throughout the study period is prohibited. Note: during the study period, opioid agonists should be avoided as they may be rendered ineffective by samidorphan.

### 8.4.3. Permitted Therapy

Permissible potential medications to treat extrapyramidal symptoms may include benzodiazepines, antihistamines, and anticholinergics. Benzodiazepines should be utilized for treatment-emergent akathisia. While insomnia may be treated with a variety of agents, short half-life benzodiazepines should be utilized due to the potential for lingering effects on daytime functioning and study assessments (eg, triazolam). Nonbenzodiazepine medication may be used to treat insomnia (eg, zolpidem, eszopiclone). Treatment of agitation and/or anxiety with benzodiazepines is permissible.

#### 8.4.4. Pain Management

Because ALKS 3831 contains samidorphan, a μ-opioid receptor antagonist, patients may experience reduced or ineffective analgesia when taking an opioid analgesic agent concurrently with ALKS 3831, including several days after last dosing of ALKS 3831.

In the event of an emergency, pain management of the subject should include the following:

- Regional analgesia or use of non-opioid analgesics
- If opiate anesthesia or analgesia is required, the subject should be continuously monitored, in an anesthesia care setting, by persons not involved in the conduct of the surgical or diagnostic procedure. The opioid therapy must be provided by individuals specifically trained in the use of anesthetic drugs and the management of the respiratory effects of potent opioids, specifically the establishment and the maintenance of a patent airway and assisted ventilation
- Close monitoring by appropriately trained personnel in a setting equipped and staffed for cardiopulmonary resuscitation

For subjects requiring emergency opioid analgesics prior to dosing, the study drug should not be administered. If opioid analgesics are required after the study drug has been dosed, it may take several days for opiate sensitivity to be restored, since samidorphan is an opioid antagonist and could interfere with opioid-mediated pain management.

## 8.4.5. Other Restrictions and Requirements

Additional restrictions and requirements include:

- Prohibited substances include amphetamines (including methamphetamine), cocaine, barbiturates, methadone, opiates (including morphine, oxycodone, methadone, and buprenorphine), and PCP
- Subjects will be required to abstain from blood or blood product donation during the study and for 30 days following the Follow-up Visit
- Subjects will be instructed to maintain their normal caffeine intake and/or tobacco use, as well as normal activity/exercise throughout the study. Subjects will be asked to abstain from strenuous physical activity for 48 hours prior to each study visit
- Subjects will be asked to refrain from driving, operating machinery, or engaging in hazardous activities until they and the Investigator are sure the study drug is not impairing their judgment and/or ability to perform skilled tasks

## 9. TREATMENT OF SUBJECTS

## 9.1. Study Drug Dose and Administration

Study drugs include:

• ALKS 3831 10/10 (10 mg olanzapine/10 mg samidorphan), 15/10 (15 mg olanzapine/10 mg samidorphan), or 20/10 (20 mg olanzapine/10 mg samidorphan) administered as a coated bilayer tablet

At Visit 1 and all subsequent visits until EOT, subjects will be given blister cards containing study drug to take at home. Subjects will be instructed to take one tablet by mouth each day, preferably at bedtime. Dosing may be switched to another time, at the Investigator's discretion, if there are tolerability problems; however, frequent switching is discouraged.

Subjects will be instructed to keep all unused tablets in their blister card and to return unused tablets to the study site at their next visit. If dosing is to occur at that visit, the dose should be taken from the subject's next blister card, not from the card they are returning.

If a dose is missed or forgotten, subjects will be instructed to resume regular dosing the following night. Subjects will be instructed not to take a double dose to try to "make up" for the missed dose

## 9.2. Treatment Adherence

Subjects will undergo a study drug adherence review at the timepoints indicated in Table 3. Subjects will be instructed to keep all unused tablets in their original containers and to return the original containers with any unused study drug at each visit following dispensation. Study drug accountability will be documented as the number of tablets dispensed, dosed, lost/missing, or remaining. If applicable, the site will discuss nonadherence with the subject.

# 9.3. Randomization/Method of Assigning Subjects to Treatment

Not applicable.

# 9.4. Blinding

Not applicable. Study is open-label.

## 10. STUDY DRUG MATERIALS AND MANAGEMENT

## 10.1. Study Drug

The ALKS 3831 drug product will be supplied as a coated bilayer tablet in three fixed-dose combinations:

- ALKS 3831 10/10 (10 mg olanzapine/10 mg samidorphan)
- ALKS 3831 15/10 (15 mg olanzapine/10 mg samidorphan)
- ALKS 3831 20/10 (20 mg olanzapine/10 mg samidorphan)

Samidorphan is a Schedule II controlled substance. Thus, ALKS 3831 should be treated as a Schedule II controlled substance in the US and any other country in which it is controlled.

## 10.2. Packaging and Labeling

ALKS 3831 will be supplied in blister packs. Blister cards will be in weekly and biweekly configurations. Weekly blister cards will contain 9 tablets, enough for 1 week of dosing, plus sufficient overage for two additional once daily doses. Biweekly blister cards will contain 16 tablets, enough for 2 weeks of dosing, plus sufficient overage for two additional once daily doses.

## 10.3. Storage

Product should be stored 15-25°C.

Under the US Controlled Substances Act, samidorphan is considered a Schedule II substance because it is derived from opium alkaloids. Therefore, ALKS 3831 must be stored in accordance with restrictions related to Schedule II substances. The site will take adequate precautions, including storage of the investigational drug in a securely locked, substantially constructed cabinet, or other securely locked, substantially constructed enclosure, access to which is limited, to prevent theft or diversion of the substance.

# 10.4. Accountability

The Investigator will be responsible for the oversight of recording the receipt and administration of study drug, and for insuring the supervision of the storage and allocation of these supplies. The Investigator is required to maintain current drug dispensing and accountability logs throughout the study. The Investigator may delegate accountability duties to an appropriate and qualified pharmacist or staff member who is under the supervision of the Investigator. The Investigator or designee must allow the Clinical Research Associate or equivalent to perform drug reconciliation during each study monitoring visit. All unused supplies will be checked against the study drug movement records before investigational drug is returned or destroyed.

Refer to Section 8.3.11 for additional study drug reconciliation procedures.

# 10.5. Handling and Disposal

Following completion and verification of accountability logs, all unused and used packages must be destroyed. Packages may be destroyed on site according to Good Clinical Practice (GCP) and site practice. Alternatively, the Sponsor may arrange for destruction with a third party vendor operating in accordance with GCP and/or Good Manufacturing Practice (GMP), as applicable.
## 11. ASSESSMENT OF EFFICACY

The following efficacy assessments will be used to analyze the durability of treatment effect:

- PANSS
- CGI-S

#### **Other Assessments:**

The following assessments will be used to obtain information regarding subject experience throughout the study:

- IWQOL-Lite
- Cigarette Use
- EQ-5D

# 12. ASSESSMENT OF PHARMACOKINETICS AND PHARMACODYNAMICS

Not applicable.

#### 13. ASSESSMENT OF SAFETY

Safety will be assessed on the basis of:

- AEs
- Clinical laboratory parameters (chemistry, hematology, and urinalysis)
- Vital signs (oral temperature, respiratory rate, orthostatic blood pressure, and pulse)
- Weight and waist circumference
- ECG parameters (heart rate, RR, PR, QRS, and QT)
- C-SSRS
- AIMS
- BARS
- SAS

#### 13.1. Definition of Adverse Event

An AE is any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product. The occurrence, which may or may not have a causal relationship with the investigational treatment, may include any clinical or laboratory change that does not commonly occur in that subject and is considered clinically significant.

Illnesses present prior to the subject signing the informed consent form (ICF) are considered to be pre-existing conditions and are documented on the medical history eCRF. Pre-existing conditions that worsen during the study are entered on the AE eCRF.

All out-of-range laboratory values will be deemed as clinically significant or not clinically significant by the Investigator. Clinically significant values will be considered AEs and recorded as such on the eCRFs.

Pregnancy is not considered an AE, although a subject will be withdrawn from the study if a pregnancy occurs. As described in Section 8.4.1, the pregnancy must be reported to Alkermes and additional follow-up may be required.

#### 13.2. Definition of Serious Adverse Event

An SAE is any AE, occurring at any dose and regardless of causality that meets one or more of the following criteria:

- Results in death
- Is life-threatening. The subject is at immediate risk of death from the reaction as it occurs. This does not include a reaction that, had it occurred in a more severe form, might have caused death
- Requires inpatient hospitalization or prolongation of existing hospitalization

- Results in persistent or significant disability/incapacity (eg, a substantial disruption of a person's ability to conduct normal life functions)
- Is a congenital anomaly/birth defect

Important medical events that may not result in death, be immediately life-threatening, or require hospitalization may be considered to be SAEs when, based upon appropriate medical judgment, they may jeopardize the patient or subject and may require intervention to prevent one of the other outcomes listed above.

Admission to a hospital or an inpatient unit for a nonmedical reason (ie, social stay admission) during the study in the absence of untoward medical occurrence will not be considered an SAE, but will be captured as an AE.

Hospitalization due to worsening of behavioral health-related issues should be reported as an SAE.

### 13.3. Relationship to Study Drug

The assessment of study drug relationship to each AE will be reported on the appropriate source document (and SAE form, in the event of an SAE) by the Investigator (or designated Subinvestigator) according to his/her best clinical judgment. The criteria listed in Table 5 should be used to guide this assessment. Please note that not all criteria must be present to be indicative of a particular drug relationship. All study drugs are considered "test drugs" for the purposes of the definitions listed in the table.

 Table 5:
 Adverse Event Causality Guidelines

| Relationship | Criteria for Assessment |
|---|---|
| Definitely related | There is evidence of exposure to the test drug. |
| | AND |
| | The temporal sequence of the AE onset relative to administration of the test drug is reasonable. |
| | The AE is more likely explained by the test drug than by another cause. |
| | Dechallenge (if performed) is positive. |
| | Rechallenge (if feasible) is positive. |
| | The AE shows a pattern consistent with previous knowledge of the test drug or test drug class. |
| Probably related | There is evidence of exposure to the test drug. |
| | AND |
| | The temporal sequence of the AE onset relative to administration of the test drug is reasonable. |
| | The AE is more likely explained by the test drug than by another cause. |
| | Dechallenge (if performed) is positive. |
| Possibly related | There is evidence of exposure to the test drug. |
| | AND |
| | The temporal sequence of the AE onset relative to administration of the test drug is reasonable. |
| | The AE could have been due to another equally likely cause. |
| | Dechallenge (if performed) is positive. |
| Probably not | There is evidence of exposure to the test drug. |
| related | AND |
| | There is another more likely cause of the AE. |
| | Dechallenge (if performed) is negative or ambiguous. |
| | Rechallenge (if performed) is negative or ambiguous. |
| Definitely not | The subject did not receive the test drug. |
| related | OR |
| | Temporal sequence of the AE onset relative to administration of the test drug is not reasonable. |
| | OR |
| | There is another obvious cause of the AE. |

Abbreviation: AE=adverse event

#### 13.4. Monitoring and Recording of Adverse Events

Adverse event data collection will begin after a subject signs the ICF and will continue until completion of the Safety Follow-up Visit (Visit 30) or 28 days after the final dose of study drug. Any AE or SAE having an onset after the Safety Follow-up Visit will not be collected or reported unless the Investigator feels that the event may be related to the study drug.

Subjects will be instructed by the Investigator or Designee to report the occurrence of any AE. All volunteered, elicited, and observed AEs are to be recorded on the AE eCRFs.

The Investigator will assess all AEs regarding any causal relationship to the study drug (see Section 13.3), the intensity (severity) of the event, action taken, and subject outcome.

The following criteria should be used to guide the assessment of intensity (severity):

- **Mild:** Causes awareness of sign or symptom, but is easily tolerated; does not interfere with usual activities
- Moderate: Causes discomfort enough to interfere with usual activities
- Severe: Is incapacitating; results in inability to work or perform usual activities

All AEs will be followed until resolution, until deemed stable by the Investigator, or until the subject is deemed by the Investigator to be lost to follow-up.

For clinical study safety reporting purposes, the most recent version of the Investigator's Brochure will be used as the reference document to designate event expectedness.

Withdrawal from the study as a result of an AE and any therapeutic measures that are taken shall be at the discretion of the Investigator. If a subject withdraws from the study <u>for any reason</u>, any ongoing AEs will be followed until resolution, until deemed stable by the Investigator, or until the subject is deemed by the Investigator to be lost to follow-up.

## 13.5. Reporting of Serious Adverse Events and Pregnancy

All SAEs and pregnancies must be reported to Alkermes via PPD Limited immediately, within 24 hours of discovery, by emailing or faxing the report to the following:



The written report for SAEs should be submitted on the SAE form provided for this purpose. The SAE report must include the Investigator's opinion as to whether the event is study drug-related. If this relationship is determined to be possibly, probably, or definitely related to study drug, evidence to support this assessment must also be provided.

The written report for pregnancies in female subjects and in female partners of male subjects should be submitted on the Pregnancy Report Form provided for this purpose.

#### 14. STATISTICS

#### **14.1.** Sample Size Considerations

No formal sample size calculation was performed for this extension study. A sample size of approximately 390 subjects is based on the estimated maximum number of subjects who might be expected to continue from the ALK3831-A305 study.

#### 14.2. General Statistical Methodology

In general, summary statistics (n, mean, standard deviation, median, minimum and maximum values for continuous variables, and number and percentage of subjects in each category for categorical variables) will be provided for evaluated variables. All individual subject level data will be presented as data listings.

The statistical analysis methods are described below. Additional details will be provided in the Statistical Analysis Plan to be finalized before database lock.

#### 14.2.1. Study Population

#### 14.2.1.1. Safety Population

The Safety Population includes all enrolled subjects who received at least one dose of ALKS 3831.

#### 14.2.1.2. Full Analysis Set

The Full Analysis Set (FAS) Population includes all enrolled subjects who received at least one dose of ALKS 3831 and underwent at least one postdose PANSS assessment.

## 14.3. Demographics and Baseline Data

Demographics and baseline characteristics, such as gender, age, race, weight, and BMI, will be summarized with descriptive statistics.

# 14.4. Safety and Tolerability Analyses

Safety analyses will be carried out using the Safety Population. Incidence of AEs will be analyzed as a safety endpoint. Reported AE terms will be coded using the Medical Dictionary for Regulatory Activities (MedDRA) and will be summarized by system organ class and preferred term categories.

Serious AEs and AEs leading to study discontinuation (AEDCs) will also be summarized.

Observed values and changes from Baseline in weight, BMI, waist circumference, laboratory parameters, vital signs, and ECG parameters will be summarized by study visit.

The number and percentage of subjects who have met potentially clinically significant (PCS) criteria at any post-Baseline visit will be summarized for laboratory, vital signs, weight, and ECG parameters. Supporting listings will be provided.

The number and percentage of subjects with shifts in laboratory and extrapyramidal symptom (EPS) parameters (AIMS, BARS, and SAS) will be summarized. Supporting listings will be provided.

The number and percentage of subjects with C-SSRS assessments of suicidal ideation and behavior will be summarized.

Prior and concomitant medication use will be summarized by World Health Organization (WHO) Drug Dictionary Anatomical Therapeutic Class (ATC) code.

Listings will be provided for all safety endpoints.

### 14.5. Efficacy Analysis

Efficacy analyses will be carried out using the FAS Population. The following endpoints will be used to evaluate durability of treatment effect:

- Change from Baseline in PANSS total score and subscales by visit
- Change from Baseline in CGI-S by visit
- PANSS response
- Relapse
- Remission
- Time to discontinuation

The PANSS (total and subscale scores) and CGI-S scores, and appropriate changes from Baseline, will be summarized using descriptive statistics. Positive and Negative Syndrome Scale response and remission at each visit will be summarized as number and percentage.

The discontinuation rate and the relapse rate will be estimated using the Kaplan-Meier (KM) Method and the KM plot will be provided.

## 14.6. Pharmacokinetic/Pharmacodynamic Analyses

Not applicable.

#### 15. DIRECT ACCESS TO SOURCE DATA/DOCUMENTS

#### 15.1. Study Monitoring

Monitoring of the study site (including, but not limited to, reviewing eCRFs for accuracy and completeness) will be performed by an Alkermes monitor or designee.

#### 15.2. Audits and Inspections

By signing the protocol, the Investigator agrees that, within local regulatory restrictions and institutional and ethical considerations, authorized representatives of Alkermes, a regulatory authority, and/or an institutional review board (IRB)/independent ethics committee (IEC) may visit the site to perform audits or inspections, including the drug storage area, study drug stocks, drug accountability records, subject charts and source documents, and other records relative to study conduct. The purpose of an Alkermes audit or inspection is to systematically and independently examine all study-related activities and documents (eg, laboratory reports, x-rays, workbooks, subject medical records) to determine whether these activities were conducted, and whether data were recorded, analyzed, and accurately reported according to the protocol, GCP guidelines of the International Council on Harmonisation (ICH), and any applicable regulatory requirements.

The Investigator should contact Alkermes immediately if contacted by a regulatory agency regarding an inspection.

## 15.3. Institutional Review Board/Independent Ethics Committee

The Investigator must obtain IRB/IEC approval for the investigation. Initial IRB/IEC approval, as well as all materials approved by the IRB/IEC for this study, including the subject consent form and recruitment materials, must be maintained by the Investigator and made available for inspection.

#### 16. QUALITY CONTROL AND QUALITY ASSURANCE

This study will be conducted under GCP and all applicable regulatory requirements. To ensure data accuracy, completeness, and compliance, the study site should have processes in place for data review and quality control. Alkermes may also conduct a quality assurance audit. Please see Section 15.2 for details regarding the audit process.

#### 16.1. Case Report Forms

This study will use eCRFs. All eCRF data must be based on source documents or approved to be the original data (ie, data directly reported on the eCRF). All eCRFs will be completed by the clinic staff prior to review by the Alkermes monitor or designated representative.

The Alkermes monitor or designated representative will review all source records on-site and compare them to the data collected on the eCRF.

#### 16.2. Confidentiality of Data

By signing this protocol, the Investigator affirms to Alkermes that he or she will maintain in confidence information furnished to him or her by Alkermes and will divulge such information to his or her respective IRB or IEC under an appropriate understanding of confidentiality with such board. All data will be considered the sole property of Alkermes. Please refer to the Clinical Study Agreement (CSA) for details.

#### 17. ETHICAL CONSIDERATIONS

#### 17.1. Ethics Review

The clinical site's IRB/IEC must meet all relevant regulatory requirements. The study protocol and ICF will be reviewed by the IRB/IEC prior to enrolling subjects into the study; written approval from the committee must be received by Alkermes before drug will be released to the Investigator. The protocol must be re-approved by the IRB/IEC upon receipt of amendments and annually, as local regulatory requirements require.

The Investigator is responsible for submitting all protocol changes and SAE reports to the IRB/IEC according to local procedures. At a minimum, all SAEs requiring an investigational new drug safety report must be immediately reported.

All relevant correspondence from the IRB/IEC will be forwarded by the respective study site to the Sponsor in a timely fashion.

#### 17.2. Ethical Conduct of the Study

This study will be conducted in accordance with the protocol, the ICH Guideline E6, and all applicable local regulatory requirements. Good Clinical Practice is an international ethical and scientific quality standard used for designing, conducting, recording, and reporting studies involving the participation of human subjects. Alkermes is committed to complying with this standard to provide assurance that the rights, safety, and well-being of study subjects will be protected, consistent with the principles having their origin in the Declaration of Helsinki.

#### 17.3. Written Informed Consent

The Investigator (or authorized designee) at each center will ensure that the subject (or the subject's legal representative) is given full and adequate oral and written information about the nature, purpose, potential and possible risks and benefits of the study. Each prospective subject will receive an IRB/IEC-approved ICF that summarizes the pertinent study information and will be given ample time to read the form and ask questions about the study. All information is to be provided in a language understandable to the subject and must not include any language that waives the subject's legal rights. Prospective subjects must also be informed of their right to withdraw consent without prejudice at any time during the study. If the subject chooses to participate, he/she must sign the ICF before any study-specific procedures are conducted.

All subjects will be informed of their rights to privacy and will be made aware that the study data will be submitted to Alkermes, the IRB/IEC, the CRO, if applicable, and to regulatory authorities for review and evaluation for the duration of the study and until the project has been approved for marketing, or is withdrawn from investigation. They will also be informed that the Study Monitor may inspect their medical records to verify the accuracy and completeness of the study records and results.

Significant changes to the protocol or product safety information may require a revision of the ICF, which must be reviewed and approved by the IRB/IEC, and then signed by all applicable study participants.

The time that informed consent is obtained must be documented. The Investigator must maintain the original, signed ICF in the subject's source documents. A copy of the signed ICF must be given to the subject.

#### 18. DATA HANDLING AND RECORDKEEPING

An overview of study data handling and recordkeeping procedures and restrictions is provided in the subsequent sections; please refer to the CSA for further details.

#### 18.1. Data Capture

As stated in Section 16.1, this study will use eCRFs for capturing data. All entries, corrections, and alterations will be made by the Investigator or other authorized study personnel. All data entries will be verified for accuracy and correctness by independent monitors. The electronic data capture system maintains a full audit trail.

All electronic source data collected outside of the eCRF, such as central laboratory data, will be transferred directly to Alkermes for incorporation into the final datasets. A paper copy of all laboratory reports will remain with the source documents at the study site. All out-of-range laboratory values will be deemed as clinically significant or not clinically significant by the Investigator. Clinically significant values will be considered AEs and recorded as such on the eCRFs.

Adverse events will be coded using the MedDRA. Concomitant medications will be categorized using the WHO-ATC classification system.

#### 18.2. Inspection of Records

Alkermes or its representative will be allowed to conduct site visits to the investigational facilities for the purpose of monitoring any aspect of the study. The Investigator agrees to allow the monitor to inspect the drug storage area, study drug stocks, drug accountability records, subject charts and source documents, and other records relative to study conduct.

#### 18.3. Retention of Records

Retention and storage of all essential clinical study documents shall be governed by the terms and conditions of the site's CSA and in accordance with ICH guidelines/local regulatory requirements as follows:

Essential documents should be retained until at least 2 years after the last approval of a marketing application in an ICH region and until there are no pending or contemplated marketing applications in an ICH region, or at least 2 years have elapsed since the formal discontinuation of clinical development of the investigational product. These documents should be retained for a longer period, however, if required by the applicable regulatory requirements or by the terms of the CSA. It is the responsibility of the Sponsor to inform the Investigator/institution as to when these documents no longer need to be retained.

Subject medical files should be retained in accordance with the applicable legislation and in accordance with the maximum period of time permitted by the hospital, institution, or private practice.

# 18.4. Use of Information and Publication Policy

Data generated in this study are proprietary information that is the sole property of Alkermes. Results of the study are to be held in confidence by both the investigators and the Sponsor.

Please refer to the CSA for details on the procedures for publishing and presenting data.

#### 19. REFERENCES

Barnes TR. A rating scale for drug-induced akathisia. *Br J Psychiatry*. 1989;154:672-676.

Dixon L. Dual diagnosis of substance abuse in schizophrenia: prevalence and impact on outcomes. *Schizophr Res.* 1999;35 Suppl:S93-100.

Zyprexa (olanzapine) [package insert]. Indianapolis, IN: Eli Lilly and Company; 2017.

Food and Drug Administration. Drug Development and Drug Interactions: Table of Substrates, Inhibitors and Inducers. 2016;

http://www.fda.gov/Drugs/DevelopmentApprovalProcess/DevelopmentResources/DrugInteractionsLabeling/ucm093664.htm. Accessed on: 18 Apr 2017.

Guy W. *ECDEU Assessment Manual for Psychopharmacology*. Rockville, MD: Department of Health, Education, and Welfare; 1976.

Harris EC, Barraclough B. Excess mortality of mental disorder. *Br J Psychiatry*. 1998;173:11-53.

Hodgins S. Violent behaviour among people with schizophrenia: a framework for investigations of causes, and effective treatment, and prevention. *Philos Trans R Soc Lond B Biol Sci.* 2008;363(1503):2505-2518. doi: 10.1098/rstb.2008.0034.

Kay S, Fiszbein A, Opler L. The Positive and Negative Syndrome Scale (PANSS) for Schizophrenia. *Schizophr Bull.* 1987;13(2):261-276.

Koekkoek B, van MB, Hutschemaekers G. "Difficult patients" in mental health care: a review. *Psychiatr Serv.* 2006;57(6):795-802. doi: 10.1176/appi.ps.57.6.795.

Kuo CJ, Tsai SY, Lo CH, Wang YP, Chen CC. Risk factors for completed suicide in schizophrenia. *J Clin Psychiatry*. 2005;66(5):579-585.

Lambert M, Conus P, Cotton S, Robinson J, McGorry PD, Schimmelmann BG. Prevalence, Predictors, and Consequences of Long-Term Refusal of Antipsychotic Treatment in First-Episode Psychosis. *J Clin Psychopharmacol.* 2010;30(5):565-572. doi: 10.1097/JCP.0b013e3181f058a0.

Lieberman JA, Stroup TS, McEvoy JP, et al. Effectiveness of antipsychotic drugs in patients with chronic schizophrenia. *N Engl J Med.* 2005;353(12):1209-1223.

Nasrallah HA, Meyer JM, Goff DC, et al. Low rates of treatment for hypertension, dyslipidemia and diabetes in schizophrenia: data from the CATIE schizophrenia trial sample at baseline. *Schizophr Res.* 2006;86(1-3):15-22. doi: 10.1016/j.schres.2006.06.026.

Posner K, Brown GK, Stanley B, et al. The Columbia-Suicide Severity Rating Scale: initial validity and internal consistency findings from three multisite studies with adolescents and adults. *Am J Psychiatry*. 2011;168(12):1266-1277. doi: 10.1176/appi.ajp.2011.10111704.

Regier DA, Farmer ME, Rae DS, et al. Comorbidity of mental disorders with alcohol and other drug abuse. Results from the Epidemiologic Catchment Area (ECA) Study. *JAMA*. 1990;264(19):2511-2518.

Saha S, Chant D, McGrath J. A systematic review of mortality in schizophrenia: is the differential mortality gap worsening over time? *Arch Gen Psychiatry*. 2007;64(10):1123-1131. doi: 10.1001/archpsyc.64.10.1123.

Simpson GM, Angus JW. A rating scale for extrapyramidal side effects. *Acta Psychiatr Scand Suppl.* 1970;212:11-19.

Tiihonen J, Lonnqvist J, Wahlbeck K, et al. 11-year follow-up of mortality in patients with schizophrenia: a population-based cohort study (FIN11 study). *Lancet*. 2009;374(9690):620-627. doi: 10.1016/S0140-6736(09)60742-X.

University of Washington: School of Pharmacy. In Vivo CYP3A Inducers. Seattle, WA: M and T Drug Interaction Database; 2017a.

University of Washington: School of Pharmacy. In Vivo Inhibitors of CYP3A Probes. Seattle, WA: M and T Drug Interaction Database; 2017b.

#### 20. APPENDICES

**Appendix A:** Partial List of Prohibited Cytochrome P450 (CYP) 3A4 Inhibitors and Inducers

**Appendix B:** Positive and Negative Syndrome Scale

**Appendix C:** Clinical Global Impression

Severity

**Appendix D:** Abnormal Involuntary Movement Scale

**Appendix E:** Barnes Akathisia Rating Scale

**Appendix F:** Simpson-Angus Scale

**Appendix G:** Columbia-Suicide Severity Rating Scale

Since Last Visit

**Appendix H:** Impact of Weight on Quality of Life-Lite

**Appendix I:** EuroQOL–5D

# APPENDIX A. PARTIAL LIST OF PROHIBITED CYTOCHROME P450 (CYP) 3A4 INHIBITORS AND INDUCERS

The following is a list of CYP3A4 inhibitors and inducers that subjects are to avoid within 30 days of Screening and throughout the study. This list is not comprehensive.

Table 1: Partial List of CYP3A4 Inhibitors and Inducers

| Moderate-to- | -Strong Inhibitors | Moderate-to-Strong Inducers |
|---|---|---|
| Aprepitant | Idelalisib | Avasimibe |
| Boceprevir | Indinavir/ Ritonavir <sup>a</sup> | Bosentan |
| Cimetidine | Itraconazole | Carbamazepine |
| Ciprofloxacin | Ketoconazole | Efavirenz |
| Clarithromycin | Lopinavir/ Ritonavir <sup>a</sup> | Enzalutamide |
| Clotrimazole | Mibefradil | Etravirine |
| Cobicistat | Nefazodone | Mitotane |
| Conivaptan | Nelfinavir | Modafinil |
| Crizotinib | Paritaprevir/ Ritonavir and (Ombitasvir and/or Dasabuvir) <sup>a</sup> | Phenobarbital |
| Cyclosporine | Posaconazole | Phenytoin |
| Danoprevir/ Ritonavir <sup>a</sup> | Ritonavir <sup>a</sup> | Rifabutin |
| Diltiazem | Saquinavir/ Ritonavir <sup>a</sup> | Rifampin |
| Dronedarone | Telaprevir | St. John's Wort |
| Elvitegravir/ Ritonavir <sup>a</sup> | Telithromycin | - |
| Erythromycin | Tipranavir/ Ritonavir <sup>a</sup> | - |
| Fluconazole | Tofisopam | - |
| Fluvoxamine | Troleandomycin | - |
| Grapefruit Juice | Verapamil | - |
| Imatinib | Voriconazole | - |

<sup>&</sup>lt;sup>a</sup> Ritonavir is usually given in combination with other anti-human immunodeficiency virus (HIV) or anti-hepatitis C virus (HCV) drugs in clinical practice. Caution should be used when extrapolating the observed effect of ritonavir alone to the effect of combination regimens on CYP3A activities.

Source: (Food and Drug Administration 2016; University of Washington: School of Pharmacy 2017a; University of Washington: School of Pharmacy 2017b)

## APPENDIX B. POSITIVE AND NEGATIVE SYNDROME SCALE



#### Positive Scale (P)

P1. Delusions. Beliefs which are unfounded, unrealistic, and idiosyncratic. Basis for rating: thought content expressed in the interview and its influence on social relations and behavior as reported by primary care workers or family.

| | Rating | Criteria |
|---|---|---|
| 1 | Absent | Definition does not apply. |
| 2 | Minimal | Questionable pathology; may be at the upper extreme of normal limits. |
| 3 | Mild | Presence of one or two delusions, which are vague, uncrystallized, and not tenaciously held. Delusions do not interfere with thinking, social relations, or behavior. |
| 4 | Moderate | Presence of either a kaleidoscopic array of poorly formed, unstable delusions or a few well-formed delusions that occasionally interfere with thinking, social relations, or behavior. |
| 5 | Moderate | Presence of numerous well-formed delusions that are tenaciously held and occasionally interfere with thinking, social relations, or behavior. |
| 6 | Severe | Presence of a stable set of delusions which are crystallized, possibly systematized, tenaciously held, and clearly interfere with thinking, social relations, and behavior. |
| 7 | Extreme | Presence of a stable set of delusions which are either highly systematized or very numerous, and which dominate major facets of the patient's life. This frequently results in inappropriate and irresponsible action, which may even jeopardize the safety of the patient or others. |

# Positive Scale (P)

P2. Conceptual disorganization. Disorganized process of thinking characterized by disruption of goal-directed sequencing, e.g., circumstantiality, tangentiality, loose associations, non-sequiturs, gross illogicality, or thought block. Basis for rating: cognitive verbal processes observed during the course of interview.

| | Rating | Criteria |
|---|---|---|
| 1 | Absent | Definition does not apply. |
| 2 | Minimal | Questionable pathology; may be at the upper extreme of normal limits. |
| 3 | Mild | Thinking is circumstantial, tangential, or paralogical. There is some difficulty in directing thoughts toward a goal, and some loosening of associations may be evidenced under pressure. |
| 4 | Moderate | Able to focus thoughts when communications are brief and structured, but becomes loose or irrelevant when dealing with more complex communications or when under minimal pressure. |
| 5 | Moderate<br>Severe | Generally has difficulty in organizing thoughts, as evidenced by frequent irrelevancies, disconnectedness, or loosening of associations even when not under pressure. |
| 6 | Severe | Thinking is seriously derailed and internally inconsistent, resulting in gross irrelevancies and disruption of thought processes, which occur almost constantly. |
| 7 | Extreme | Thoughts are disrupted to the point where the patient is incoherent. There is marked loosening of associations, which results in total failure of communication, e.g., "word salad" or mutism. |

#### Positive Scale (P)

P3. Hallucinatory behavior. Verbal report or behavior indicating perceptions which are not generated by external stimuli. These may occur in the auditory, visual, olfactory, or somatic realms. Basis for rating: verbal report and physical manifestations during the course of interview as well as reports of behavior by primary care workers or family.

| | Rating | Criteria |
|---|---|---|
| 1 | Absent | Definition does not apply. |
| 2 | Minimal | Questionable pathology; may be at the upper extreme of normal limits. |
| 3 | Mild | One or two clearly formed but infrequent hallucinations, or else a number of vague abnormal perceptions, which do not result in distortions of thinking or behavior. |
| 4 | Moderate | Hallucinations occur frequently but not continuously, and the patient's thinking and behavior are affected only to a minor extent. |
| 5 | Moderate<br>Severe | Hallucinations are frequent, may involve more than one sensory modality, and tend to distort thinking and/or disrupt behavior. Patient may have delusional interpretation of these experiences and respond to them emotionally and, on occasion, verbally as well. |
| 6 | Severe | Hallucinations are present almost continuously, causing major disruption of thinking and behavior. Patient treats these as real perceptions, and functioning is impeded by frequent emotional and verbal responses to them. |
| 7 | Extreme | Patient is almost totally preoccupied with hallucinations, which virtually dominate thinking and behavior. Hallucinations are provided a rigid delusional interpretation and provoke verbal and behavioral responses, including obedience to command hallucinations. |

# Positive Scale (P)

P4. Excitement. Hyperactivity as reflected in accelerated motor behavior, heightened responsivity to stimuli, hypervigilance, or excessive mood lability. Basis for rating: behavioral manifestations during the course of interview as well as reports of behavior by primary care workers or family.

| | Rating | Criteria |
|---|---|---|
| 1 | Absent | Definition does not apply. |
| 2 | Minimal | Questionable pathology; may be at the upper extreme of normal limits. |
| 3 | Mild | Tends to be slightly agitated, hypervigilant, or mildly overaroused throughout the interview, but without distinct episodes of excitement or marked mood lability. Speech may be slightly pressured. |
| 4 < | Moderate | Agitation or overarousal is clearly evident throughout the interview, affecting speech and general mobility, or episodic outbursts occur sporadically. |
| 5 | Moderate<br>Severe | Significant hyperactivity or frequent outbursts of motor activity are observed, making it difficult for the patient to sit still for longer than several minutes at any given time. |
| 6 | Severe | Marked excitement dominates the interview, delimits attention, and to some extent affects personal functions such as eating and sleeping. |
| 7 | Extreme | Marked excitement seriously interferes in eating and sleeping and makes interpersonal interactions virtually impossible. Acceleration of speech and motor activity may result in incoherence and exhaustion. |

#### Positive Scale (P)

**P5.** Grandiosity. Exaggerated self-opinion and unrealistic convictions of superiority, including delusions of extraordinary abilities, wealth, knowledge, fame, power, and moral righteousness. Basis for rating: thought content expressed in the interview and its influence on behavior as reported by primary care workers or family.

| | Rating | Criteria |
|---|---|---|
| 1 | Absent | Definition does not apply. |
| 2 | Minimal | Questionable pathology; may be at the upper extreme of normal limits. |
| 3 | Mild | Some expansiveness or boastfulness is evident, but without clear-cut grandiose delusions. |
| 4 | Moderate | Feels distinctly and unrealistically superior to others. Some poorly formed delusions about special status or abilities may be present but are not acted upon. |
| 5 | Moderate<br>Severe | Clear-cut delusions concerning remarkable abilities, status, or power are expressed and influence attitude but not behavior. |
| 6 | Severe | Clear-cut delusions of remarkable superiority involving more than one parameter (wealth, knowledge, fame, etc.) are expressed, notably influence interactions, and may be acted upon. |
| 7 | Extreme | Thinking, interactions, and behavior are dominated by multiple delusions of amazing ability, wealth, knowledge, fame, power, and/or moral stature, which may take on a bizarre quality. |

## Positive Scale (P)

**P6.** Suspiciousness/persecution. Unrealistic or exaggerated ideas of persecution, as reflected in guardedness, a distrustful attitude, suspicious hypervigilance, or frank delusions that others mean one harm. Basis for rating: thought content expressed in the interview and its influence on behavior as reported by primary care workers or family.

| | Rating | Criteria |
|---|---|---|
| 1 | Absent | Definition does not apply. |
| 2 | Minimal | Questionable pathology; may be at the upper extreme of normal limits. |
| 3 | Mild | Presents a guarded or even openly distrustful attitude, but thoughts, interactions, and behavior are minimally affected. |
| 4 | Moderate | Distrustfulness is clearly evident and intrudes on the interview and/or behavior, but there is no evidence of persecutory delusions. Alternatively, there may be indication of loosely formed persecutory delusions, but these do not seem to affect the patient's attitude or interpersonal relations. |
| 5 | Moderate<br>Severe | Patient shows marked distrustfulness, leading to major disruption of interpersonal relations, or else there are clear-cut persecutory delusions that have limited impact on interpersonal relations and behavior. |
| 6 | Severe | Clear-cut pervasive delusions of persecution which may be systematized and significantly interfere in interpersonal relations. |
| 7 | Extreme | A network of systematized persecutory delusions dominates the patient's thinking, social relations, and behavior. |

#### Positive Scale (P)

P7. Hostility. Verbal and nonverbal expressions of anger and resentment, including sarcasm, passive-aggressive behavior, verbal abuse, and assaultiveness. Basis for rating: interpersonal behavior observed during the interview and reports by primary care workers or family.

| | Rating | Criteria |
|---|---|---|
| 1 | Absent | Definition does not apply. |
| 2 | Minimal | Questionable pathology; may be at the upper extreme of normal limits. |
| 3 | Mild | Indirect or restrained communication of anger, such as sarcasm, disrespect, hostile expressions, and occasional irritability. |
| 4 | Moderate | Presents an overtly hostile attitude, showing frequent irritability and direct expression of anger or resentment. |
| 5 | Moderate<br>Severe | Patient is highly irritable and occasionally verbally abusive or threatening. |
| 6 | Severe | Uncooperativeness and verbal abuse or threats notably influence the interview and seriously impact upon social relations. Patient may be violent and destructive but is not physically assaultive toward others. |
| 7 | Extreme | Marked anger results in extreme uncooperativeness, precluding other interactions, or in episode(s) of physical assault toward others. |

# Negative Scale (N)

N1. Blunted affect. Diminished emotional responsiveness as characterized by a reduction in facial expression, modulation of feelings, and communicative gestures. Basis for rating: observation of physical manifestations of affective tone and emotional responsiveness during the course of interview.

| | Rating | Criteria |
|---|---|---|
| 1 | Absent | Definition does not apply. |
| 2 | Minimal | Questionable pathology; may be at the upper extreme of normal limits. |
| 3 | Mild | Changes in facial expression and communicative gestures seem to be stilted, forced, artificial, or lacking in modulation. |
| 4 | Moderate | Reduced range of facial expression and few expressive gestures result in a dull appearance. |
| 5 | Moderate<br>Severe | Affect is generally "flat," with only occasional changes in facial expression and a paucity of communicative gestures. |
| 6 | Severe | Marked flatness and deficiency of emotions exhibited most of the time. There may be unmodulated extreme affective discharges, such as excitement, rage, or inappropriate uncontrolled laughter. |
| 7 | Extreme | Changes in facial expression and evidence of communicative gestures are virtually absent. Patient seems constantly to show a barren or 'wooden' expression. |

#### Negative Scale (N)

N2. Emotional withdrawal. Lack of interest in, involvement with, and affective commitment to life's events. Basis for rating: reports of functioning from primary care workers or family and observation of interpersonal behavior during the course of interview.

| | Rating | Criteria |
|---|---|---|
| 1 | Absent | Definition does not apply. |
| 2 | Minimal | Questionable pathology; may be at the upper extreme of normal limits. |
| 3 | Mild | Usually lacks initiative and occasionally may show deficient interest in surrounding events. |
| 4 | Moderate | Patient is generally distanced emotionally from the milieu and its challenges but, with encouragement, can be engaged. |
| 5 | Moderate<br>Severe | Patient is clearly detached emotionally from persons and events in the milieu, resisting all efforts at engagement. Patient appears distant, docile, and purposeless but can be involved in communication at least briefly and tends to personal needs, sometimes with assistance. |
| 6 | Severe | Marked deficiency of interest and emotional commitment results in limited conversation with others and frequent neglect of personal functions, for which the patient requires supervision. |
| 7 | Extreme | Patient is almost totally withdrawn, uncommunicative, and neglectful of personal needs as a result of profound lack of interest and emotional commitment. |

# Negative Scale (N)

N3. Poor rapport. Lack of interpersonal empathy, openness in conversation, and sense of closeness, interest, or involvement with the interviewer. This is evidenced by interpersonal distancing and reduced verbal and nonverbal communication. Basis for rating: interpersonal behavior during the course of interview.

| | Rating | Criteria |
|---|---|---|
| 1 | Absent | Definition does not apply. |
| 2 | Minimal | Questionable pathology; may be at the upper extreme of normal limits. |
| 3 | Mild | Conversation is characterized by a stilted, strained, or artificial tone. It may lack emotional depth or tend to remain on an impersonal, intellectual plane. |
| 4 | Moderate | Patient typically is aloof, with interpersonal distance quite evident. Patient may answer questions mechanically, act bored, or express disinterest. |
| 5 | Moderate<br>Severe | Disinvolvement is obvious and clearly impedes the productivity of the interview. Patient may tend to avoid eye or face contact. |
| 6 | Severe | Patient is highly indifferent, with marked interpersonal distance. Answers are perfunctory, and there is little nonverbal evidence of involvement. Eye and face contact are frequently avoided. |
| 7 | Extreme | Patient is totally uninvolved with the interviewer. Patient appears to be completely indifferent and consistently avoids verbal and nonverbal interactions during the interview. |

#### Negative Scale (N)

N4. Passive/apathetic social withdrawal. Diminished interest and initiative in social interactions due to passivity, apathy, anergy, or avolition. This leads to reduced interpersonal involvements and neglect of activities of daily living. Basis for rating: reports on social behavior from primary care workers or family.

| | Rating | Criteria |
|---|---|---|
| 1 | Absent | Definition does not apply. |
| 2 | Minimal | Questionable pathology; may be at the upper extreme of normal limits. |
| 3 | Mild | Shows occasional interest in social activities but poor initiative. Usually engages with others only when approached first by them. |
| 4 | Moderate | Passively goes along with most social activities but in a disinterested or mechanical way. Tends to recede into the background. |
| 5 | Moderate<br>Severe | Passively participates in only a minority of activities and shows virtually no interest or initiative. Generally spends little time with others. |
| 6 | Severe | Tends to be apathetic and isolated, participating very rarely in social activities and occasionally neglecting personal needs. Has very few spontaneous social contacts. |
| 7 | Extreme | Profoundly apathetic, socially isolated, and personally neglectful. |

# Negative Scale (N)

N5. Difficulty in abstract thinking. Impairment in the use of the abstract-symbolic mode of thinking, as evidenced by difficulty in classification, forming generalizations, and proceeding beyond concrete or egocentric thinking in problem-solving tasks. Basis for rating: responses to questions on similarities and proverb interpretation, and use of concrete vs. abstract mode during the course of the interview.

| | Rating | Criteria |
|---|---|---|
| 1 | Absent | Definition does not apply. |
| 2 | Minimal | Questionable pathology; may be at the upper extreme of normal limits. |
| 3 | Mild | Tends to give literal or personalized interpretations to the more difficult proverbs and may have some problems with concepts that are fairly abstract or remotely related. |
| 4 | Moderate | Often utilizes a concrete mode. Has difficulty with most proverbs and some categories. Tends to be distracted by functional aspects and salient features. |
| 5 | Moderate<br>Severe | Deals primarily in a concrete mode, exhibiting difficulty with most proverbs and many categories. |
| 6 | Severe | Unable to grasp the abstract meaning of any proverbs or figurative expressions and can formulate classifications for only the most simple of similarities. Thinking is either vacuous or locked into functional aspects, salient features, and idiosyncratic interpretations. |
| 7 | Extreme | Can use only concrete modes of thinking. Shows no comprehension of proverbs, common metaphors or similes, and simple categories. Even salient and functional attributes do not serve as a basis for classification. This rating may apply to those who cannot interact even minimally with the examiner due to marked cognitive impairment. |

#### Negative Scale (N)

N6. Lack of spontaneity and flow of conversation. Reduction in the normal flow of communication associated with apathy, avolition, defensiveness, or cognitive deficit. This is manifested by diminished fluidity and productivity of the verbal-interactional process. Basis for rating: cognitive-verbal processes observed during the course of interview.

| | Rating | Criteria |
|---|---|---|
| 1 | Absent | Definition does not apply. |
| 2 | Minimal | Questionable pathology; may be at the upper extreme of normal limits. |
| 3 | Mild | Conversation shows little initiative. Patient's answers tend to be brief and unembellished, requiring direct and leading questions by the interviewer. |
| 4 | Moderate | Conversation lacks free flow and appears uneven or halting. Leading questions are frequently needed to elicit adequate responses and proceed with conversation. |
| 5 | Moderate<br>Severe | Patient shows a marked lack of spontaneity and openness, replying to the interviewer's questions with only one or two brief sentences. |
| 6 | Severe | Patient's responses are limited mainly to a few words or short phrases intended to avoid or curtail communication. (E.g., "I don't know," "I'm not at liberty to say.") Conversation is seriously impaired as a result, and the interview is highly unproductive. |
| 7 | Extreme | Verbal output is restricted to, at most, an occasional utterance, making conversation impossible. |

## Negative Scale (N)

N7. Stereotyped thinking. Decreased fluidity, spontaneity, and flexibility of thinking, as evidenced in rigid, repetitious, or barren thought content. Basis for rating: cognitive-verbal processes observed during the interview.

| | Rating | Criteria |
|---|---|---|
| 1 | Absent | Definition does not apply. |
| 2 | Minimal | Questionable pathology; may be at the upper extreme of normal limits. |
| 3 | Mild | Some rigidity shown in attitudes or beliefs. Patient may refuse to consider alternative positions or have difficulty in shifting from one idea to another. |
| 4 | Moderate | Conversation revolves around a recurrent theme, resulting in difficulty in shifting to a new topic. |
| 5 | Moderate<br>Severe | Thinking is rigid and repetitious to the point that, despite the interviewer's efforts, conversation is limited to only two or three dominating topics. |
| 6 | Severe | Uncontrolled repetition of demands, statements, ideas, or questions which severely impairs conversation. |
| 7 | Extreme | Thinking, behavior, and conversation are dominated by constant repetition of fixed ideas or limited phrases, leading to gross rigidity, inappropriateness, and restrictiveness of patient's communication. |

#### General Psychopathology Scale (G)

G1. Somatic concern. Physical complaints or beliefs about bodily illness or malfunctions. This may range from a vague sense of ill being to clear-cut delusions of catastrophic physical disease. Basis for rating: thought content expressed in the interview.

| | Rating | Criteria |
|---|---|---|
| 1 | Absent | Definition does not apply. |
| 2 | Minimal | Questionable pathology; may be at the upper extreme of normal limits. |
| 3 | Mild | Distinctly concerned about health or somatic issues, as evidenced by occasional questions and desire for reassurance. |
| 4 | Moderate | Complains about poor health or bodily malfunction, but there is no delusional conviction, and over-concern can be allayed by reassurance. |
| 5 | Moderate<br>Severe | Patient expresses numerous or frequent complaints about physical illness or bodily malfunction, or else patient reveals one or two clear-cut delusions involving these themes but is not preoccupied by them. |
| 6 | Severe | Patient is preoccupied by one or a few clear-cut delusions about physical disease or organic malfunction, but affect is not fully immersed in these themes, and thoughts can be diverted by the interviewer with some effort. |
| 7 | Extreme | Numerous and frequently reported somatic delusions, or only a few somatic delusions of a catastrophic nature, which totally dominate the patient's affect and thinking. |

## General Psychopathology Scale (G)

G2. Anxiety. Subjective experience of nervousness, worry, apprehension, or restlessness, ranging from excessive concern about the present or future to feelings of panic. Basis for rating: verbal report during the course of interview and corresponding physical manifestations.

| | Rating | Criteria |
|---|---|---|
| 1 | Absent | Definition does not apply. |
| 2 | Minimal | Questionable pathology; may be at the upper extreme of normal limits. |
| 3 | Mild | Expresses some worry, over-concern, or subjective restlessness, but no somatic and behavioral consequences are reported or evidenced. |
| 4 | Moderate | Patient reports distinct symptoms of nervousness, which are reflected in mild physical manifestations such as fine hand tremor and excessive perspiration. |
| 5 | Moderate<br>Severe | Patient reports serious problems of anxiety, which have significant physical and behavioral consequences, such as marked tension, poor concentration, palpitations, or impaired sleep. |
| 6 | Severe | Subjective state of almost constant fear associated with phobias, marked restlessness, or numerous somatic manifestations. |
| 7 | Extreme | Patient's life is seriously disrupted by anxiety, which is present almost constantly and, at times, reaches panic proportion or is manifested in actual panic attacks. |

#### General Psychopathology Scale (G)

G3. Guilt feelings. Sense of remorse or self-blame for real or imagined misdeeds in the past. Basis for rating: verbal report of guilt feelings during the course of interview and the influence on attitudes and thoughts.

| | Rating | Criteria |
|---|---|---|
| 1 | Absent | Definition does not apply. |
| 2 | Minimal | Questionable pathology; may be at the upper extreme of normal limits. |
| 3 | Mild | Questioning elicits a vague sense of guilt or self-blame for a minor incident, but the patient clearly is not overly concerned. |
| 4 | Moderate | Patient expresses distinct concern over his or her responsibility for a real incident in his or her life but is not preoccupied with it, and attitude and behavior are essentially unaffected. |
| 5 | Moderate<br>Severe | Patient expresses a strong sense of guilt associated with self-deprecation or the belief that he or she deserves punishment. The guilt feelings may have a delusional basis, may be volunteered spontaneously, may be a source of preoccupation and/or depressed mood, and cannot be allayed readily by the interviewer. |
| 6 | Severe | Strong ideas of guilt take on a delusional quality and lead to an attitude of hopelessness or worthlessness. The patient believes he or she should receive harsh sanctions for the misdeeds and may even regard his or her current life situation as such punishment. |
| 7 | Extreme | Patient's life is dominated by unstable delusions of guilt, for which he or she feels deserving of drastic punishment, such as life imprisonment, torture, or death. There may be associated suicidal thoughts or attribution of others' problems to one's own past misdeeds. |

# General Psychopathology Scale (G)

G4. Tension. Overt physical manifestations of fear, anxiety, and agitation, such as stiffness, tremor, profuse sweating, and restlessness. Basis for rating: verbal report attesting to anxiety and, thereupon, the severity of physical manifestations of tension observed during the interview.

| | Rating | Criteria |
|---|---|---|
| 1 | Absent | Definition does not apply. |
| 2 | Minimal | Questionable pathology; may be at the upper extreme of normal limits. |
| 3 | Mild | Posture and movements indicate slight apprehensiveness, such as minor rigidity, occasional restlessness, shifting of position, or fine rapid hand tremor. |
| 4 | Moderate | A clearly nervous appearance emerges from various manifestations, such as fidgety behavior, obvious hand tremor, excessive perspiration, or nervous mannerisms. |
| 5 | Moderate<br>Severe | Pronounced tension is evidenced by numerous manifestations, such as nervous shaking, profuse sweating, and restlessness, but conduct in the interview is not significantly affected. |
| 6 | Severe | Pronounced tension to the point that interpersonal interactions are disrupted. The patient, for example, may be constantly fidgeting, unable to sit still for long, or show hyperventilation. |
| 7 | Extreme | Marked tension is manifested by signs of panic or gross motor acceleration, such as rapid restless pacing and inability to remain seated for longer than a minute, which makes sustained conversation not possible. |

#### General Psychopathology Scale (G)

G5. Mannerisms and posturing. Unnatural movements or posture as characterized by an awkward, stilted, disorganized, or bizarre appearance. Basis for rating: observation of physical manifestations during the course of interview as well as reports from primary care workers or family.

| | Rating | Criteria |
|---|---|---|
| 1 | Absent | Definition does not apply. |
| 2 | Minimal | Questionable pathology; may be at the upper extreme of normal limits. |
| 3 | Mild | Slight awkwardness in movements or minor rigidity of posture. |
| 4 | Moderate | Movements are notably awkward or disjointed, or an unnatural posture is maintained for brief periods. |
| 5 | Moderate<br>Severe | Occasional bizarre rituals or contorted posture are observed, or an abnormal position is sustained for extended periods. |
| 6 | Severe | Frequent repetition of bizarre rituals, mannerisms, or stereotyped movements, or a contorted posture is sustained for extended periods. |
| 7 | Extreme | Functioning is seriously impaired by virtually constant involvement in ritualistic, manneristic, or stereotyped movements or by an unnatural fixed posture which is sustained most of the time. |

# General Psychopathology Scale (G)

G6. Depression. Feelings of sadness, discouragement, helplessness, and pessimism. Basis for rating: verbal report of depressed mood during the course of interview and its observed influence on attitude and behavior as reported by primary care workers or family.

| | Rating | Criteria |
|---|---|---|
| 1 | Absent | Definition does not apply. |
| 2 | Minimal | Questionable pathology; may be at the upper extreme of normal limits. |
| 3 | Mild | Expresses some sadness or discouragement only on questioning, but there is no evidence of depression in general attitude or demeanor. |
| 4 | Moderate | Distinct feelings of sadness or hopelessness, which may be spontaneously divulged, but depressed mood has no major impact on behavior or social functioning, and the patient usually can be cheered up. |
| 5 | Moderate<br>Severe | Distinctly depressed mood is associated with obvious sadness, pessimism, loss of social interest, psychomotor retardation, and some interference in appetite and sleep. The patient cannot be easily cheered up. |
| 6 | Severe | Markedly depressed mood is associated with sustained feelings of misery, occasional crying, hopelessness, and worthlessness. In addition, there is major interference in appetite and/or sleep as well as in normal motor and social functions, with possible signs of self-neglect. |
| 7 | Extreme | Depressive feelings seriously interfere in most major functions. The manifestations include frequent crying, pronounced somatic symptoms, impaired concentration, psychomotor retardation, social disinterest, self-neglect, possible depressive or nihilistic delusions, and/or possible suicidal thoughts or actions. |

#### General Psychopathology Scale (G)

G7. Motor retardation. Reduction in motor activity as reflected in slowing or lessening of movements and speech, diminished responsiveness to stimuli, and reduced body tone. Basis for rating: manifestations during the course of interview as well as reports by primary care workers or family.

| | Rating | Criteria |
|---|---|---|
| 1 | Absent | Definition does not apply. |
| 2 | Minimal | Questionable pathology; may be at the upper extreme of normal limits. |
| 3 | Mild | Slight but noticeable diminution in rate of movements and speech. Patient may be somewhat underproductive in conversation and gestures. |
| 4 | Moderate | Patient is clearly slow in movements, and speech may be characterized by poor productivity, including long response latency, extended pauses, or slow pace. |
| 5 | Moderate<br>Severe | A marked reduction in motor activity renders communication highly unproductive or delimits functioning in social and occupational situations. Patient can usually be found sitting or lying down. |
| 6 | Severe | Movements are extremely slow, resulting in a minimum of activity and speech. Essentially the day is spent sitting idly or lying down. |
| 7 | Extreme | Patient is almost completely immobile and virtually unresponsive to external stimuli. |

# General Psychopathology Scale (G)

G8. Uncooperativeness. Active refusal to comply with the will of significant others, including the interviewer, hospital staff, or family, which may be associated with distrust, defensiveness, stubbornness, negativism, rejection of authority, hostility, or belligerence. Basis for rating: interpersonal behavior observed during the course of interview as well as reports by primary care workers or family.

| | Rating | Criteria |
|---|---|---|
| 1 | Absent | Definition does not apply. |
| 2 | Minimal | Questionable pathology; may be at the upper extreme of normal limits. |
| 3 | Mild | Complies with an attitude of resentment, impatience, or sarcasm. May inoffensively object to sensitive probing during the interview. |
| 4 | Moderate | Occasional outright refusal to comply with normal social demands, such as making own bed, attending scheduled programs, etc. The patient may project a hostile, defensive, or negative attitude but usually can be worked with. |
| 5 | Moderate<br>Severe | Patient frequently is incompliant with the demands of his or her milieu and may be characterized by others as an "outcast' or having "a serious attitude problem." Uncooperativeness is reflected in obvious defensiveness or irritability with the interviewer and possible unwillingness to address many questions. |
| 6 | Severe | Patient is highly uncooperative, negativistic, and possibly also belligerent. Refuses to comply with most social demands and may be unwilling to initiate or conclude the full interview. |
| 7 | Extreme | Active resistance seriously impacts on virtually all major areas of functioning. Patient may refuse to join in any social activities, tend to personal hygiene, converse with family or staff, and participate even briefly in an interview. |

#### General Psychopathology Scale (G)

G9. Unusual thought content. Thinking characterized by strange, fantastic, or bizarre ideas, ranging from those, which are remote or atypical to those which are distorted, illogical, and patently absurd. Basis for rating: thought content expressed during the course of interview.

| | Rating | Criteria |
|---|---|---|
| 1 | Absent | Definition does not apply. |
| 2 | Minimal | Questionable pathology; may be at the upper extreme of normal limits. |
| 3 | Mild | Thought content is somewhat peculiar or idiosyncratic, or familiar ideas are framed in an odd context. |
| 4 | Moderate | Ideas are frequently distorted and occasionally seem quite bizarre. |
| 5 | Moderate<br>Severe | Patient expresses many strange and fantastic thoughts (e.g., being the adopted son of a king, being an escapee from death row) or some which are patently absurd (e.g., having hundreds of children, receiving radio messages from outer space through a tooth filling). |
| 6 | Severe | Patient expresses many illogical or absurd ideas or some, which have a distinctly bizarre quality (e.g., having three heads, being a visitor from another planet). |
| 7 | Extreme | Thinking is replete with absurd, bizarre, and grotesque ideas. |

## General Psychopathology Scale (G)

G10. Disorientation. Lack of awareness of one's relationship to the milieu, including persons, place, and time, which may be due to confusion or withdrawal. Basis for rating: responses to interview questions on orientation.

| | Rating | Criteria |
|---|---|---|
| 1 | Absent | Definition does not apply. |
| 2 | Minimal | Questionable pathology; may be at the upper extreme of normal limits. |
| 3 | Mild | General orientation is adequate but there is some difficulty with specifics. For example, patient knows his or her location but not the street address; knows hospital staff names but not their functions; knows the month but confuses the day of week with an adjacent day; or errs in the date by more than two days. There may be narrowing of interest evidenced by familiarity with the immediate but not extended milieu, such as ability to identify staff but not the Mayor, Governor, or President. |
| 4 | Moderate | Only partial success in recognizing persons, places, and time. For example, patient knows he or she is in a hospital but not its name; knows the name of his or her city but not the borough or district, knows the name of his or her primary therapist but not many other direct care workers; knows the year and season but is not sure of the month. |
| 5 | Moderate<br>Severe | Considerable failure in recognizing persons, place, and time. Patient has only a vague notion of where he or she is and seems unfamiliar with most people in his or her milieu. He or she may identify the year correctly or nearly so but not know the current month, day of week, or even the season. |
| 6 | Severe | Marked failure in recognizing persons, place, and time. For example, patient has no knowledge of his or her whereabouts; confuses the date by more than one year; can name only one or two individuals in his or her current life. |
| 7 | Extreme | Patient appears completely disoriented with regard to persons, place, and time. There is gross confusion or total ignorance about one's location, the current year, and even the most familiar people, such as parents, spouse, friends, and primary therapist. |

#### General Psychopathology Scale (G)

G11. Poor attention. Failure in focused alertness manifested by poor concentration, distractibility from internal and external stimuli, and difficulty in harnessing, sustaining, or shifting focus to new stimuli. Basis for rating: manifestations during the course of interview.

| | Rating | Criteria |
|---|---|---|
| 1 | Absent | Definition does not apply. |
| 2 | Minimal | Questionable pathology; may be at the upper extreme of normal limits. |
| 3 | Mild | Limited concentration evidenced by occasional vulnerability to distraction or faltering attention toward the end of the interview. |
| 4 | Moderate | Conversation is affected by the tendency to be easily distracted, difficulty in long sustaining concentration on a given topic, or problems in shifting attention to new topics. |
| 5 | Moderate<br>Severe | Conversation is seriously hampered by poor concentration, distractibility, and difficulty in shifting focus appropriately. |
| 6 | Severe | Patient's attention can be harnessed for only brief moments or with great effort, due to marked distraction by internal or external stimuli. |
| 7 | Extreme | Attention is so disrupted that even brief conversation is not possible. |

# General Psychopathology Scale (G)

G12. Lack of judgment and insight. Impaired awareness or understanding of one's own psychiatric condition and life situation. This is evidenced by failure to recognize past or present psychiatric illness or symptoms, denial of need for psychiatric hospitalization or treatment, decisions characterized by poor anticipation of consequences, and unrealistic short-term and long-range planning. Basis for rating: thought content expressed during the interview.

| | Rating | Criteria |
|---|---|---|
| 1 | Absent | Definition does not apply. |
| 2 | Minimal | Questionable pathology; may be at the upper extreme of normal limits. |
| 3 | Mild | Recognizes having a psychiatric disorder but clearly underestimates its seriousness, the implications for treatment, or the importance of taking measures to avoid relapse. Future planning may be poorly conceived. |
| 4 | Moderate | Patient shows only a vague or shallow recognition of illness. There may be fluctuations in acknowledgment of being ill or little awareness of major symptoms, which are present, such as delusions, disorganized thinking, suspiciousness, and social withdrawal. The patient may rationalize the need for treatment in terms of its relieving lesser symptoms, such as anxiety, tension, and sleep difficulty. |
| 5 | Moderate<br>Severe | Acknowledges past but not present psychiatric disorder. If challenged, the patient may concede the presence of some unrelated or insignificant symptoms, which tend to be explained away by gross misinterpretation or delusional thinking. The need for psychiatric treatment similarly goes unrecognized. |
| 6 | Severe | Patient denies ever having had a psychiatric disorder. He or she disavows the presence of any psychiatric symptoms in the past or present and, though compliant, denies the need for treatment and hospitalization. |
| 7 | Extreme | Emphatic denial of past and present psychiatric illness. Current hospitalization and treatment are given a delusional interpretation (e.g., as punishment for misdeeds, as persecution by tormentors, etc.), and the patient may thus refuse to cooperate with therapists, medication, or other aspects of treatment. |

## General Psychopathology Scale (G)

G13. Disturbance of volition. Disturbance in the willful initiation, sustenance, and control of one's thoughts, behavior, movements, and speech. Basis for rating: thought content and behavior manifested in the course of interview.

| | Rating | Criteria |
|---|---|---|
| 1 | Absent | Definition does not apply. |
| 2 | Minimal | Questionable pathology; may be at the upper extreme of normal limits. |
| 3 | Mild | There is evidence of some indecisiveness in conversation and thinking, which may impede verbal and cognitive processes to a minor extent. |
| 4 | Moderate | Patient is often ambivalent and shows clear difficulty in reaching decisions. Conversation may be marred by alteration in thinking, and in consequence verbal and cognitive functioning are clearly impaired. |
| 5 | Moderate<br>Severe | Disturbance of volition interferes in thinking as well as behavior. Patient shows pronounced indecision that impedes the initiation and continuation of social and motor activities, and which also may be evidenced in halting speech. |
| 6 | Severe | Disturbance of volition interferes in the execution of simple, automatic motor functions, such as dressing and grooming, and markedly affects speech. |
| 7 | Extreme | Almost complete failure of volition is manifested by gross inhibition of movement and speech, resulting in immobility and/or mutism. |

# General Psychopathology Scale (G)

G14. Poor impulse control. Disordered regulation and control of action on inner urges, resulting in sudden, unmodulated, arbitrary, or misdirected discharge of tension and emotions without concern about consequences. Basis for rating: behavior during the course of interview and reported by primary care workers or family.

| | Rating | Criteria |
|---|---|---|
| 1 | Absent | Definition does not apply. |
| 2 | Minimal | Questionable pathology; may be at the upper extreme of normal limits. |
| 3 | Mild | Patient tends to be easily angered and frustrated when facing stress or denied gratification but rarely acts on impulse. |
| 4 | Moderate | Patient gets angered and verbally abusive with minimal provocation. May be occasionally threatening, destructive, or have one or two episodes involving physical confrontation or a minor brawl. |
| 5 | Moderate<br>Severe | Patient exhibits repeated impulsive episodes involving verbal abuse, destruction of property, or physical threats. There may be one or two episodes involving serious assault, for which the patient requires isolation, physical restraint, or p.r.n. sedation. |
| 6 | Severe | Patient frequently is impulsively aggressive, threatening, demanding, and destructive, without any apparent consideration of consequences. Shows assaultive behavior and may also be sexually offensive and possibly respond behaviorally to hallucinatory commands. |
| 7 | Extreme | Patient exhibits homicidal attacks, sexual assaults, repeated brutality, or self-destructive behavior. Requires constant direct supervision or external constraints because of inability to control dangerous impulses. |

## General Psychopathology Scale (G)

G15. Preoccupation. Absorption with internally generated thoughts and feelings and with autistic experiences to the detriment of reality orientation and adaptive behavior. Basis for rating: interpersonal behavior observed during the course of interview.

| | Rating | Criteria |
|---|---|---|
| 1 | Absent | Definition does not apply. |
| 2 | Minimal | Questionable pathology; may be at the upper extreme of normal limits. |
| 3 | Mild | Excessive involvement with personal needs or problems, such that conversation veers back to egocentric themes and there is diminished concern exhibited toward others. |
| 4 | Moderate | Patient occasionally appears self-absorbed, as if daydreaming or involved with internal experiences, which interferes with communication to a minor extent. |
| 5 | Moderate<br>Severe | Patient often appears to be engaged in autistic experiences, as evidenced by behaviors that significantly intrude on social and communicational functions, such as the presence of a vacant stare, muttering or talking to oneself, or involvement with stereotyped motor patterns. |
| 6 | Severe | Marked preoccupation with autistic experiences, which seriously delimits concentration, ability to converse, and orientation to the milieu. The patient frequently may be observed smiling, laughing, muttering, talking, or shouting to himself or herself. |
| 7 | Extreme | Gross absorption with autistic experiences, which profoundly affects all major realms of behavior. The patient constantly may be responding verbally and behaviorally to hallucinations and show little awareness of other people or the external milieu. |

# General Psychopathology Scale (G)

G16. Active social avoidance. Diminished social involvement associated with unwarranted fear, hostility, or distrust. Basis for rating: reports of social functioning by primary care workers or family.

| | Rating | Criteria |
|---|---|---|
| 1 | Absent | Definition does not apply. |
| 2 | Minimal | Questionable pathology; may be at the upper extreme of normal limits. |
| 3 | Mild | Patient seems ill at ease in the presence of others and prefers to spend time alone, although he or she participates in social functions when required. |
| 4 | Moderate | Patient grudgingly attends all or most social activities but may need to be persuaded or may terminate prematurely on account of anxiety, suspiciousness, or hostility. |
| 5 | Moderate<br>Severe | Patient fearfully or angrily keeps away from many social interactions despite others' efforts to engage him. Tends to spend unstructured time alone. |
| 6 | Severe | Patient participates in very few social activities because of fear, hostility, or distrust. When approached, the patient shows a strong tendency to break off interactions, and generally he or she appears to isolate himself or herself from others. |
| 7 | Extreme | Patient cannot be engaged in social activities because of pronounced fears, hostility, or persecutory delusions. To the extent possible, he or she avoids all interactions and remains isolated from others. |
# APPENDIX C. CLINICAL GLOBAL IMPRESSION

• Severity

# Clinical Global Impressions- Severity

| Name or ID: | Date: |
|----------------|-------|
| Trainio di IBI | |

Instructions: Circle the appropriate number after the following item.

#### **SEVERITY OF ILLNESS**

Considering your total clinical experience with this particular population, how mentally ill is the patient at this time?

- 0 Not assessed
- 1 Normal, not at all ill
- 2 Borderline mentally ill
- 3 Mildly ill
- 4 Moderately ill
- 5 Markedly ill
- 6 Severely ill
- 7 Among the most extremely ill patients

This tool should be used to supplement, not to replace, clinical judgement.

## APPENDIX D. ABNORMAL INVOLUNTARY MOVEMENT SCALE

#### Abnormal Involuntary Movement Scale (AIMS)

| • | Rate highest severity observed. Rate movements that occur upon activation observed spontaneously. | Code:<br>0 = Non<br>1 = Mini<br>2 = Mild<br>3 = Mod<br>4 = Seve | mal, ma<br>erate | y be extr | eme no | rmal | | |
|---|---|---|---|---|---|---|---|---|
| | | | | | (Circle | One) | | |
| | MUSCLES OF FACIAL EXPRESSION e.g movements of forehead, eyeb periorbital area, cheeks, including frowning, blinking, smiling, grimacing | orows, | 0 | 1 | 2 | 3 | 4 | |
| FACIAL AND<br>ORAL | 2. LIPS AND PERIORAL AREA e.g. puckering, pouting, smacking | | 0 | 1 | 2 | 3 | 4 | |
| MOVEMENTS: | 3. JAW e.g. biting, clenching, chewing, mouth opening, lateral movement | | 0 | 1 | 2 | 3 | 4 | |
| | 4. TONGUE Rate only increases in movement both in and out of mouth. NO inability to sustain movement | DΤ | 0 | 1 | 2 | 3 | 4 | |
| EXTREMITY<br>MOVEMENTS: | <ol> <li>UPPER (ARMS, WRISTS, HANDS, FINGERS) Include choreic movemen<br/>rapid, objectively purposeless, irregular, spontaneous), athetoid movemer<br/>slow, irregular, complex, serpentine). Do NOT include tremor (i.e. repetitive<br/>regular, rhythmic)</li> </ol> | nts (i.e. | 0 | 1 | 2 | 3 | 4 | |
| | 6. LOWER (LEGS, KNEES, ANKLES, TOES) e.g. lateral knee movement, f tapping, heel dropping, foot squirming, inversion and eversion of foot | foot | 0 | 1 | 2 | 3 | 4 | |
| TRUNK<br>MOVEMENTS: | 7. NECK, SHOULDERS, HIPS e.g.rocking, twisting, squirming, pelvic gyratic | ions | 0 | 1 | 2 | 3 | 4 | |
| | 8. SEVERITY OF ABNORMAL MOVEMENTS | | | | N | None, norr<br>Minir<br>N<br>Moder<br>Sev | nal 1<br>lild 2<br>ate 3 | 0<br>1<br>2<br>3<br>4 |
| GLOBAL<br>JUDGMENT: | 9. INCAPACITATION DUE TO ABNORMAL MOVEMENTS | | | | N | None, norr<br>Minir<br>N<br>Moder<br>Sev | nal 1<br>lild 2<br>ate 3 | 0<br>1<br>2<br>3<br>4 |
| | 10. PATIENT'S AWARENESS OF ABNORMAL MOVEMENTS. RATE ONL | Υ | | | | | | , |
| | PATIENT'S REPORT | | | | | o awarene | | 0 |
| | | | | | | e, no distre<br>mild distre | | 1<br>2 |
| | | | | | , | rniid distre | | 3 |
| | | | | | • | vere distre | | 4 |
| | 11. Current problems with teeth and/or dentures? | | | | | | | 0 |
| DENTAL | | | | | | | Yes 1 | |
| STATUS: | 12. Does patient usually wear dentures? | | | | | | No ( | 0 |
| | | | | | | , | Yes 1 | 1 |

| Rater Signature: | Date: |
|------------------|-------|
| Natel Signature. | Date. |

## APPENDIX E. BARNES AKATHISIA RATING SCALE

#### Barnes Akathisia Rating Scale (BARS)

**Instructions:** Patient should be observed while they are seated, and then standing while engaged in neutral conversation (for a minimum of two minutes in each position). Symptoms observed in other situations, for example, while engaged in activity on the ward, may also be rated. Subsequently, the subjective phenomena should be elicited by direct questioning. **Please circle the appropriate scores.** 

#### **Objective**

- **0** Normal, occasional fidgety movements of the limbs
- Presence of characteristic restless movements: shuffling or tramping movements of the legs/feet, or swinging of one leg while sitting, *and/or* rocking from foot to foot or "walking on the spot" when standing, *but* movements present for less than half the time observed
- 2 Observed phenomena, as described in (1) above, which are present for at least half the observation period
- Patient is constantly engaged in characteristic restless movements, *and/or* has the inability to remain seated or standing without walking or pacing, during the time observed

#### Subjective

Awareness of restlessness

- 0 Absence of inner restlessness
- 1 Non-specific sense of inner restlessness
- 2 The patient is aware of an inability to keep the legs still, or a desire to move the legs, *and/or* complains of inner restlessness aggravated specifically by being required to stand still
- 3 Awareness of an intense compulsion to move most of the time and/or reports strong desire to walk or pace most of the time

Distress related to restlessness

- 0 No distress
- 1 Mild
- 2 Moderate
- 3 Severe

#### **Global Clinical Assessment of Akathisia**

- Absent. No evidence of awareness of restlessness. Observation of characteristic movements of akathisia in the absence of a subjective report of inner restlessness or compulsive desire to move the legs should be classified as pseudoakathisia
- 1 Questionable. Non-specific inner tension and fidgety movements
- 2 Mild akathisia. Awareness of restlessness in the legs and/or inner restlessness worse when required to stand still. Fidgety movements present, but characteristic restless movements of akathisia not necessarily observed. Condition causes little or no distress
- Moderate akathisia. Awareness of restlessness as described for mild akathisia above, combined with characteristic restless movements such as rocking from foot to foot when standing. Patient finds the condition distressing
- 4 Marked akathisia. Subjective experience of restlessness includes a compulsive desire to walk or pace.
  However, the patient is able to remain seated for at least five minutes. The condition is obviously distressing.
- 5 Severe akathisia. The patient reports a strong compulsion to pace up and down most of the time. Unable to sit or lie down for more than a few minutes. Constant restlessness which is associated with intense distress and insomnia.

| Rater Signature: | Date: |
|------------------|-------|

#### Scoring the Barnes Akathisia Rating Scale (BARS)

The Barnes Akathisia Rating Scale is scored as follows:

Objective Akathisia, Subjective Awareness of Restlessness and Subjective Distress Related to Restlessness are rated on a 4-point scale from 0-3 and are summed yielding a total score ranging from 0 to 9.

The Global Clinical Assessment of Akathisia uses a 5-point scale ranging from 0 – 4.

Reproduced from: Barnes TR: A Rating Scale for Drug-Induced Akathisia. British Journal of Psychiatry 154:672-676, 1989.

Clintara Version 1.6 June, 2011

# APPENDIX F. SIMPSON-ANGUS SCALE

#### SIMPSON ANGUS RATING SCALE

#### Circle the appropriate score for each item:

# 1. GAIT The patient is examined as he walks into the examining room: his gait, the swing of arms, his

The patient is examined as he walks into the examining room: his gait, the swing of arms, his general posture; all form the basis for an overall score for this item. This is rated as follows:

- 0 Normal
- 1 Mild diminution in swing while the patient is walking
- 2 Obvious diminution in swing suggesting shoulder rigidity
- 3 Stiff gait with little or no arm swing noticeable
- 4 Rigid gait with arms slightly pronated; or stopped-shuffling gait with propulsion and retropulsion

#### 2. ARM DROPPING

The patient and the examiner both raise their arms to shoulder height and let them fall to their sides. In a normal subject a stout slap is heard as the arms hit the sides. In the patient with extreme Parkinson's syndrome, the arms fall very slowly.

- 0 Normal, free fall with loud slap and rebound
- 1 Fall slowed slightly with less audible contact and little rebound
- 2 Fall slowed, no rebound
- 3 Marked slowing, no slap at all
- 4 Arms fall as though against resistance; as though through glue

#### 3. SHOULDER SHAKING

The subject's arms are bent at a right angle at the elbow and are taken one at a time by the examiner who grabs one hand and also clasps the other around the patient's elbow. The subject's upper arm is pushed to and fro and the humerus is externally rotated. The degree of resistance from normal to extreme rigidity is scored as follows:

- 0 Normal
- 1 Slight stiffness and resistance
- 2 Moderate stiffness and resistance
- 3 Marked rigidity with difficulty in passive movement
- 4 Extreme stiffness and rigidity with almost a frozen joint

Modified from: Simpson GM, Angus JWS: A rating scale for extrapyramidal side effects. Acta Psychiatrica Scandinavica 212:11-19, 1970. Revised

#### 4. **ELBOW RIGIDITY** The elbow joints are separately bent at right angles and passively extended and flexed, with the subject's biceps observed and simultaneously palpated. The resistance to this procedure is rated. (The presence of cogwheel rigidity is noted separately.) 0 Normal 1 Slight stiffness and resistance 2 Moderate stiffness and resistance 3 Marked rigidity with difficulty in passive movement 4 Extreme stiffness and rigidity with almost a frozen joint 5. WRIST RIGIDITY OR FIXATION OF POSITION The wrist is held in one hand and then the fingers held by the examiner's other hand with the wrist moved to extension, and both ulnar and radial deviation. The resistance to this procedure is rated: 0 Normal 1 Slight stiffness and resistance 2 Moderate stiffness and resistance 3 Marked rigidity with difficulty in passive movement 4 Extreme stiffness and rigidity with almost a frozen joint 6. **LEG PENDULOUSNESS** The patient sits on a table with his legs hanging down and swinging free. The ankle is grasped by the examiner and raised until the knee is partially extended. It is then allowed to fall. The resistance to falling and the lack of swinging form the basis for the score on this item: 0 The legs swing freely 1 Slight diminution in the swing of the legs 2 Moderate resistance to swing 3 Marked resistance and damping of swing 4 Complete absence of swing 7. **HEAD ROTATION** The patient sits or stands and is told that you are going to move his head side to side, that it will not hurt and that he should try and relax. (Questions about pain in the cervical area or difficulty in moving his head should be obtained to avoid causing any pain.) Clasp the patient's head between the two hands with fingers on back of the neck. Gently rotate the head in a circular motion 3 times and evaluate the muscular resistance to the movement. 0 Loose, no resistance 1 Slight resistance to movement although the time to rotate may be normal 2 Resistance is apparent and time of rotation is slowed 3 Resistance is obvious and rotation is slowed Head appears stiff and rotation is difficult to carry out

| Subject ID No | Visit No |
|------------------------------|-------------------------------------------|
| Modified from: Simpson GM, | Angus JWS: A rating scale for |
| extrapyramidal side effects. | Acta Psychiatrica Scandinavica 212:11-19, |
| 1970. Revised | |

Clintara Version 1.6 June, 2011

| 8. | | <b>GLABELLA TAP</b> Subject is told to open his eyes and not to blink. The glabella region is tapped at a steady, rapid speed. The number of times patient blinks in succession is noted: |
|---|---|---|
| | 0 | 0-5 blinks |
| | 1 | 6-10 blinks |
| | 2 | 11-15 blinks |
| | 3 | 16-20 blinks |
| | 4 | 21 and more blinks |
| 9. | | TREMOR Patient is observed walking into examining room and then is examined for this item: |
| | 0 | Normal |
| | 1 | Mild finger tremor, obvious to sight and touch |
| | 2 | Tremor of hand or arm occurring spasmodically |
| | 3 | Persistent tremor of one or more limbs |
| | 4 | Whole body tremor |
| 10. | | SALIVATION Patient is observed while talking and then asked to open his mouth and elevate his tongue. The following ratings are given: |
| | 0 | Normal |
| | 1 | Excess salivation so that pooling takes place if the mouth is open and the tongue raised |
| | 2 | Excess salivation is present and might occasionally result in difficulty in speaking |
| | 3 | Speaking with difficulty because of excess salivation |
| | 4 | Frank drooling |

| Rater Signature: | Date: |
|------------------|-------|

| Subject ID No | Visit No |
|---------------|----------|
|---------------|----------|

## APPENDIX G. COLUMBIA-SUICIDE SEVERITY RATING SCALE

• Since Last Visit Version

# COLUMBIA-SUICIDE SEVERITY RATING SCALE

(C-SSRS)

Since Last Visit

Version 1/14/09

Posner, K.; Brent, D.; Lucas, C.; Gould, M.; Stanley, B.; Brown, G.; Fisher, P.; Zelazny, J.; Burke, A.; Oquendo, M.; Mann, J.

#### Disclaimer:

This scale is intended for use by trained clinicians. The questions contained in the Columbia-Suicide Severity Rating Scale are suggested probes. Ultimately, the determination of the presence of suicidality depends on clinical judgment.

Definitions of behavioral suicidal events in this scale are based on those used in **The Columbia Suicide History Form**, developed by John Mann, MD and Maria Oquendo, MD, Conte Center for the Neuroscience of Mental Disorders (CCNMD), New York State Psychiatric Institute, 1051 Riverside Drive, New York, NY, 10032. (Oquendo M. A., Halberstam B. & Mann J. J., Risk factors for suicidal behavior: utility and limitations of research instruments. In M.B. First [Ed.] Standardized Evaluation in Clinical Practice, pp. 103-130, 2003.)

For reprints of the C-SSRS contact PPD New York State Psychiatric Institute, 1051 Riverside Drive, New York, New York, 10032; inquiries and training requirements contact PPD

| SUICIDAL IDEATION | | | |
|---|---|---|---|
| | Suicidal Behavior" section. If the answer to question 2 is "yes," or 2 is "yes", complete "Intensity of Ideation" section below. | | e Last<br>isit |
| 1. Wish to be Dead Subject endorses thoughts about a wish to be dead or not alive anymore, Have you wished you were dead or wished you could go to sleep and no | | Yes | No |
| If yes, describe: | | | |
| 2. Non-Specific Active Suicidal Thoughts General, non-specific thoughts of wanting to end one's life/commit suici oneself/associated methods, intent, or plan during the assessment period. Have you actually had any thoughts of killing yourself? | de (e.g. "I've thought about killing myself") without thoughts of ways to kill | Yes | No |
| If yes, describe: | | | |
| place or method details worked out (e.g. thought of method to kill self b overdose but I never made a specific plan as to when, where or how I wo Have you been thinking about how you might do this? | nod during the assessment period. This is different than a specific plan with time, ut not a specific plan). Includes person who would say, "I thought about taking an | Yes | No |
| If yes, describe: | | | |
| 4. Active Suicidal Ideation with Some Intent to Act, withe Active suicidal thoughts of killing oneself and subject reports having som definitely will not do anything about them". Have you had these thoughts and had some intention of acting on them If yes, describe: | me intent to act on such thoughts, as opposed to "I have the thoughts but I | Yes | No |
| 5. Active Suicidal Ideation with Specific Plan and Intent Thoughts of killing oneself with details of plan fully or partially worked Have you started to work out or worked out the details of how to kill you | | Yes | No |
| If yes, describe: | | | |
| INTENSITY OF IDEATION | · | | |
| INTENSITY OF IDEATION The following features should be rated with respect to the most s and 5 being the most severe ). | severe type of ideation (i.e.,1-5 from above, with 1 being the least severe | M | ost |
| The following features should be rated with respect to the most s | severe type of ideation (i.e.,1-5 from above, with 1 being the least severe | | ost<br>⁄ere |
| The following features should be rated with respect to the most s and 5 being the most severe ). Most Severe Ideation: Type # (1-5) | nevere type of ideation (i.e.,1-5 from above, with 1 being the least severe Description of Ideation | | |
| The following features should be rated with respect to the most s and 5 being the most severe ). Most Severe Ideation: | Description of Ideation | | |
| The following features should be rated with respect to the most s and 5 being the most severe ). Most Severe Ideation: Type # (1-5) Frequency How many times have you had these thoughts? (1) Less than once a week (2) Once a week (3) 2-5 times in week Duration | Description of Ideation | | |
| The following features should be rated with respect to the most s and 5 being the most severe ). Most Severe Ideation: Type # (1-5) Frequency How many times have you had these thoughts? (1) Less than once a week (2) Once a week (3) 2-5 times in week | Description of Ideation | | |
| The following features should be rated with respect to the most s and 5 being the most severe ). Most Severe Ideation: Type # (1-5) Frequency How many times have you had these thoughts? (1) Less than once a week (2) Once a week (3) 2-5 times in wee Duration When you have the thoughts, how long do they last? (1) Fleeting - few seconds or minutes (2) Less than 1 hour/some of the time (3) 1-4 hours/a lot of time Controllability | Description of Ideation ek (4) Daily or almost daily (5) Many times each day (4) 4-8 hours/most of day (5) More than 8 hours/persistent or continuous | | |
| The following features should be rated with respect to the most s and 5 being the most severe ). Most Severe Ideation: Type # (1-5) Frequency How many times have you had these thoughts? (1) Less than once a week (2) Once a week (3) 2-5 times in wee Duration When you have the thoughts, how long do they last? (1) Fleeting - few seconds or minutes (2) Less than 1 hour/some of the time (3) 1-4 hours/a lot of time | Description of Ideation ek (4) Daily or almost daily (5) Many times each day (4) 4-8 hours/most of day (5) More than 8 hours/persistent or continuous | | |
| The following features should be rated with respect to the most s and 5 being the most severe ). Most Severe Ideation: Type # (1-5) Frequency How many times have you had these thoughts? (1) Less than once a week (2) Once a week (3) 2-5 times in wee Duration When you have the thoughts, how long do they last? (1) Fleeting - few seconds or minutes (2) Less than 1 hour/some of the time (3) 1-4 hours/a lot of time Controllability Could /can you stop thinking about killing yourself or wants (1) Easily able to control thoughts (2) Can control thoughts with little difficulty (3) Can control thoughts with some difficulty Deterrents | Description of Ideation ek (4) Daily or almost daily (5) Many times each day (4) 4-8 hours/most of day (5) More than 8 hours/persistent or continuous ing to die if you want to? (4) Can control thoughts with a lot of difficulty (5) Unable to control thoughts (0) Does not attempt to control thoughts | | |
| The following features should be rated with respect to the most s and 5 being the most severe ). Most Severe Ideation: Type # (1-5) Frequency How many times have you had these thoughts? (1) Less than once a week (2) Once a week (3) 2-5 times in wee Duration When you have the thoughts, how long do they last? (1) Fleeting - few seconds or minutes (2) Less than 1 hour/some of the time (3) 1-4 hours/a lot of time Controllability Could /can you stop thinking about killing yourself or wants (1) Easily able to control thoughts (2) Can control thoughts with little difficulty (3) Can control thoughts with some difficulty Deterrents Are there things - anyone or anything (e.g. family, religion, thoughts of committing suicide? (1) Deterrents definitely stopped you from attempting suicide | Description of Ideation ek (4) Daily or almost daily (5) Many times each day (4) 4-8 hours/most of day (5) More than 8 hours/persistent or continuous ing to die if you want to? (4) Can control thoughts with a lot of difficulty (5) Unable to control thoughts (0) Does not attempt to control thoughts pain of death) - that stopped you from wanting to die or acting on (4) Deterrents most likely did not stop you | | |
| The following features should be rated with respect to the most s and 5 being the most severe ). Most Severe Ideation: Type # (1-5) Frequency How many times have you had these thoughts? (1) Less than once a week (2) Once a week (3) 2-5 times in wee Duration When you have the thoughts, how long do they last? (1) Fleeting - few seconds or minutes (2) Less than 1 hour/some of the time (3) 1-4 hours/a lot of time Controllability Could /can you stop thinking about killing yourself or wants (1) Easily able to control thoughts (2) Can control thoughts with little difficulty (3) Can control thoughts with some difficulty Deterrents Are there things - anyone or anything (e.g. family, religion, thoughts of committing suicide? | Description of Ideation ek (4) Daily or almost daily (5) Many times each day (4) 4-8 hours/most of day (5) More than 8 hours/persistent or continuous ing to die if you want to? (4) Can control thoughts with a lot of difficulty (5) Unable to control thoughts (0) Does not attempt to control thoughts pain of death) - that stopped you from wanting to die or acting on | | |
| The following features should be rated with respect to the most s and 5 being the most severe ). Most Severe Ideation: Type # (1-5) Frequency How many times have you had these thoughts? (1) Less than once a week (2) Once a week (3) 2-5 times in wee Duration When you have the thoughts, how long do they last? (1) Fleeting - few seconds or minutes (2) Less than 1 hour/some of the time (3) 1-4 hours/a lot of time Controllability Could /can you stop thinking about killing yourself or wants (1) Easily able to control thoughts (2) Can control thoughts with little difficulty (3) Can control thoughts with some difficulty (3) Can control thoughts with some difficulty Deterrents Are there things - anyone or anything (e.g. family, religion, thoughts of committing suicide? (1) Deterrents definitely stopped you from attempting suicide (2) Deterrents probably stopped you (3) Uncertain that deterrents stopped you Reasons for Ideation What sort of reasons did you have for thinking about wanting | Description of Ideation ek (4) Daily or almost daily (5) Many times each day (4) 4-8 hours/most of day (5) More than 8 hours/persistent or continuous ing to die if you want to? (4) Can control thoughts with a lot of difficulty (5) Unable to control thoughts (0) Does not attempt to control thoughts pain of death) - that stopped you from wanting to die or acting on (4) Deterrents most likely did not stop you (5) Deterrents definitely did not stop you (6) Does not apply ing to die or killing yourself? Was it to end the pain or stop the way | | |
| The following features should be rated with respect to the most s and 5 being the most severe ). Most Severe Ideation: Type # (1-5) Frequency How many times have you had these thoughts? (1) Less than once a week (2) Once a week (3) 2-5 times in wee Duration When you have the thoughts, how long do they last? (1) Fleeting - few seconds or minutes (2) Less than 1 hour/some of the time (3) 1-4 hours/a lot of time Controllability Could /can you stop thinking about killing yourself or wants (1) Easily able to control thoughts (2) Can control thoughts with little difficulty (3) Can control thoughts with some difficulty (3) Can control thoughts with some difficulty Deterrents Are there things - anyone or anything (e.g. family, religion, thoughts of committing suicide? (1) Deterrents definitely stopped you from attempting suicide (2) Deterrents probably stopped you (3) Uncertain that deterrents stopped you Reasons for Ideation What sort of reasons did you have for thinking about wanting | Description of Ideation ek (4) Daily or almost daily (5) Many times each day (4) 4-8 hours/most of day (5) More than 8 hours/persistent or continuous ing to die if you want to? (4) Can control thoughts with a lot of difficulty (5) Unable to control thoughts (0) Does not attempt to control thoughts pain of death) - that stopped you from wanting to die or acting on (4) Deterrents most likely did not stop you (5) Deterrents definitely did not stop you (0) Does not apply | | |

| SUICIDAL BEHAVIOR | Since Last | i |
|---|---|---|
| (Check all that apply, so long as these are separate events; must ask about all types) | Visit | |
| Actual Attempt: A potentially self-injurious act committed with at least some wish to die, as a result of act. Behavior was in part thought of as method to kill oneself. Intent | Yes No | |
| does not have to be 100%. If there is <i>any</i> intent/desire to die associated with the act, then it can be considered an actual suicide attempt. <i>There does not</i> | | |
| have to be any injury or harm, just the potential for injury or harm. If person pulls trigger while gun is in mouth but gun is broken so no injury results, | | |
| this is considered an attempt. | | |
| Inferring Intent: Even if an individual denies intent/wish to die, it may be inferred clinically from the behavior or circumstances. For example, a highly lethal act that is clearly not an accident so no other intent but suicide can be inferred (e.g. gunshot to head, jumping from window of a high floor/story). | | |
| Also, if someone denies intent to die, but they thought that what they did could be lethal, intent may be inferred. | | |
| Have you made a suicide attempt? | | |
| Have you done anything to harm yourself? | | |
| Have you done anything dangerous where you could have died? | Total # of<br>Attempts | |
| What did you do? | rttempts | |
| Did you as a way to end your life? | | |
| Did you want to die (even a little) when you? Were you trying to end your life when you? | | |
| Or did you think it was possible you could have died from? | | |
| Or did you do it purely for other reasons / without ANY intention of killing yourself (like to relieve stress, feel better, get | | |
| sympathy, or get something else to happen)? (Self-Injurious Behavior without suicidal intent) | | |
| If yes, describe: | | |
| | Yes No | |
| Has subject engaged in Non-Suicidal Self-Injurious Behavior? | | |
| Interrupted Attempt: | | _ |
| When the person is interrupted (by an outside circumstance) from starting the potentially self-injurious act (if not for that, actual attempt would have occurred). | Yes No | |
| Overdose: Person has pills in hand but is stopped from ingesting. Once they ingest any pills, this becomes an attempt rather than an interrupted attempt. | | |
| Shooting: Person has gun pointed toward self, gun is taken away by someone else, or is somehow prevented from pulling trigger. Once they pull the trigger, | | |
| even if the gun fails to fire, it is an attempt. Jumping: Person is poised to jump, is grabbed and taken down from ledge. Hanging: Person has noose around neck but has not yet started to hang - is stopped from doing so. | | |
| Has there been a time when you started to do something to end your life but someone or something stopped you before you | Total # of interrupted | |
| actually did anything? | merrupica | |
| If yes, describe: | | |
| Aborted Attempt: | | _ |
| When person begins to take steps toward making a suicide attempt, but stops themselves before they actually have engaged in any self-destructive behavior. | Yes No | |
| Examples are similar to interrupted attempts, except that the individual stops him/herself, instead of being stopped by something else. | | |
| Has there been a time when you started to do something to try to end your life but you stopped yourself before you | Total # of | |
| actually did anything? If yes, describe: | aborted | |
| ii yes, describe. | | |
| Preparatory Acts or Behavior: | | _ |
| Acts or preparation towards imminently making a suicide attempt. This can include anything beyond a verbalization or thought, such as assembling a | Yes No | |
| specific method (e.g. buying pills, purchasing a gun) or preparing for one's death by suicide (e.g. giving things away, writing a suicide note). | | |
| Have you taken any steps towards making a suicide attempt or preparing to kill yourself (such as collecting pills, getting a gun, giving valuables away or writing a suicide note)? | | |
| If yes, describe: | | |
| Suicidal Behavior: | Yes No | |
| Suicidal behavior was present during the assessment period? | | |
| Completed Suicide: | Yes No | _ |
| Answer for Actual Attempts Only | Most Lethal | |
| | Attempt<br>Date: | |
| Actual Lethality/Medical Damage: | Enter Code | _ |
| 0. No physical damage or very minor physical damage (e.g. surface scratches). | Liner Couc | |
| <ol> <li>Minor physical damage (e.g. lethargic speech; first-degree burns; mild bleeding; sprains).</li> <li>Moderate physical damage; medical attention needed (e.g. conscious but sleepy, somewhat responsive; second-degree burns; bleeding of major vessel).</li> </ol> | | |
| 2. Moderately severe physical damage; medical hospitalization and likely intensive care required (e.g. comatose with reflexes intact; third-degree burns less | | |
| than 20% of body; extensive blood loss but can recover; major fractures). | | |
| 4. Severe physical damage; medical hospitalization with intensive care required (e.g. comatose without reflexes; third-degree burns over 20% of body; extensive blood loss with unstable vital signs; major damage to a vital area). | | |
| <ul><li>5. Death</li></ul> | | |
| Potential Lethality: Only Answer if Actual Lethality=0 | Enter Code | |
| Likely lethality of actual attempt if no medical damage (the following examples, while having no actual medical damage, had potential for very serious | | |
| lethality: put gun in mouth and pulled the trigger but gun fails to fire so no medical damage; laying on train tracks with oncoming train but pulled away before run over). | | |
| 0 = Behavior not likely to result in injury 1 = Behavior likely to result in injury but not likely to cause death | | |
| 2 = Behavior likely to result in death despite available medical care | | |

# APPENDIX H. IMPACT OF WEIGHT ON QUALITY OF LIFE - LITE

### Impact of Weight on Quality of Life Questionnaire—Lite Version (IWQOL-Lite)

Please answer the following statements by circling the number that best applies to you in the past week. Be as open as possible. There are no right or wrong answers.

| Phy | ysical Function | ALWAYS<br>TRUE | USUALLY<br>TRUE | SOMETIMES<br>TRUE | RARELY<br>TRUE | NEVER<br>TRUE |
|---|---|---|---|---|---|---|
| 1. | Because of my weight I have trouble picking up objects. | 5 | 4 | 3 | 2 | 1 |
| 2. | Because of my weight I have trouble tying my shoes. | 5 | 4 | 3 | 2 | 1 |
| 3. | Because of my weight I have difficulty getting up from chairs. | 5 | 4 | 3 | 2 | 1 |
| 4. | Because of my weight I have trouble using stairs. | 5 | 4 | 3 | 2 | 1 |
| 5. | Because of my weight I have difficulty putting on or taking off my clothing. | 5 | 4 | 3 | 2 | 1 |
| 6. | Because of my weight I have trouble with mobility. | 5 | 4 | 3 | 2 | 1 |
| 7. | Because of my weight I have trouble crossing my legs. | 5 | 4 | 3 | 2 | 1 |
| 8. | I feel short of breath with only mild exertion. | 5 | 4 | 3 | 2 | 1 |
| 9. | I am troubled by painful or stiff joints. | 5 | 4 | 3 | 2 | 1 |
| 10. | My ankles and lower legs are swollen at the end of the day. | 5 | 4 | 3 | 2 | 1 |
| 11. | I am worried about my health. | 5 | 4 | 3 | 2 | 1 |
| Sel | <u>f-esteem</u> | ALWAYS<br>TRUE | USUALLY<br>TRUE | SOMETIMES<br>TRUE | RARELY<br>TRUE | NEVER<br>TRUE |
| 1. | Because of my weight I am self-conscious. | 5 | 4 | 3 | 2 | 1 |
| 2. | Because of my weight my self-esteem is not what it could be. | 5 | 4 | 3 | 2 | 1 |
| 3. | Because of my weight I feel unsure of myself. | 5 | 4 | 3 | 2 | 1 |
| 4. | Because of my weight I don't like myself. | 5 | 4 | 3 | 2 | 1 |
| 5. | Because of my weight I am afraid of being rejected. | 5 | 4 | 3 | 2 | 1 |
| 6. | Because of my weight I avoid looking in mirrors or seeing myself in photographs. | 5 | 4 | 3 | 2 | 1 |
| 7. | Because of my weight I am embarrassed to be seen in public places. | 5 | 4 | 3 | 2 | 1 |

© Copyright 2000. Duke University Medical Center. Direct all correspondence to PPD Obesity and Quality of Life Consulting, 1004 Norwood Avenue, Durham, NC 27707, USA; PPD Fax: PPD

| Sex | cual Life | ALWAYS<br>TRUE | USUALLY<br>TRUE | SOMETIMES<br>TRUE | RARELY<br>TRUE | NEVER<br>TRUE |
|---|---|---|---|---|---|---|
| 1. | Because of my weight I do not enjoy sexual activity. | 5 | 4 | 3 | 2 | 1 |
| 2. | Because of my weight I have little or no sexual desire. | 5 | 4 | 3 | 2 | 1 |
| 3. | Because of my weight I have difficulty with sexual performance. | 5 | 4 | 3 | 2 | 1 |
| 4. | Because of my weight I avoid sexual encounters whenever possible. | 5 | 4 | 3 | 2 | 1 |

| Public Distress | | ALWAYS<br>TRUE | USUALLY<br>TRUE | SOMETIMES<br>TRUE | RARELY<br>TRUE | NEVER<br>TRUE |
|---|---|---|---|---|---|---|
| 1. | Because of my weight I experience ridicule, teasing, or unwanted attention. | 5 | 4 | 3 | 2 | 1 |
| 2. | Because of my weight I worry about fitting into seats in public places (e.g. theaters, restaurants, cars, or airplanes). | 5 | 4 | 3 | 2 | 1 |
| 3. | Because of my weight I worry about fitting through aisles or turnstiles. | 5 | 4 | 3 | 2 | 1 |
| 4. | Because of my weight I worry about finding chairs that are strong enough to hold my weight. | 5 | 4 | 3 | 2 | 1 |
| 5. | Because of my weight I experience discrimination by others. | 5 | 4 | 3 | 2 | 1 |
| Work (Note: For homemakers and retirees, answer with respect to your daily activities.) | | ALWAYS<br>TRUE | USUALLY<br>TRUE | SOMETIMES<br>TRUE | RARELY<br>TRUE | NEVER<br>TRUE |
| 1. | Because of my weight I have trouble getting things accomplished or meeting my responsibilities. | 5 | 4 | 3 | 2 | 1 |
| 2. | Because of my weight I am less productive than I could be. | 5 | 4 | 3 | 2 | 1 |
| 3. | Because of my weight I don't receive appropriate raises, promotions or recognition at work. | 5 | 4 | 3 | 2 | 1 |
| 4. | Because of my weight I am afraid to go on job interviews. | 5 | 4 | 3 | 2 | 1 |

© Copyright 2000. Duke University Medical Center. Direct all correspondence to PPD Obesity and Quality of Life Consulting, 1004 Norwood Avenue, Durham, NC 27707, USA; PPD Fax: PPD

# APPENDIX I. EUROQOL-5D



**Health Questionnaire** 

English version for the USA

| MOBILITY |
|---|
| I have no problems walking |
| I have slight problems walking |
| I have moderate problems walking |
| I have severe problems walking |
| I am unable to walk |
| SELF-CARE |
| I have no problems washing or dressing myself |
| I have slight problems washing or dressing myself |
| I have moderate problems washing or dressing myself |
| I have severe problems washing or dressing myself |
| I am unable to wash or dress myself |
| USUAL ACTIVITIES (e.g. work, study, housework, family or leisure activities) |
| I have no problems doing my usual activities |
| I have slight problems doing my usual activities |
| I have moderate problems doing my usual activities |
| I have severe problems doing my usual activities |
| I am unable to do my usual activities |
| PAIN / DISCOMFORT |
| I have no pain or discomfort |
| I have slight pain or discomfort |
| I have moderate pain or discomfort |
| I have severe pain or discomfort |
| I have extreme pain or discomfort |
| ANXIETY / DEPRESSION |
| I am not anxious or depressed |
| I am slightly anxious or depressed |
| I am moderately anxious or depressed |
| I am severely anxious or depressed |
| I am extremely anxious or depressed |

Under each heading, please check the ONE box that best describes your health TODAY.

The best health you can imagine

100

- 60 55
- 50 45
- 40
- 35 - 30
- 25 - 20
- 20 15 - 10

5

The worst health you can imagine

• We would like to know how good or bad your health is TODAY.

- This scale is numbered from 0 to 100.
- 100 means the <u>best</u> health you can imagine.
   0 means the <u>worst</u> health you can imagine.
- Mark an X on the scale to indicate how your health is TODAY.
- Now, please write the number you marked on the scale in the box below.

YOUR HEALTH TODAY =